

#### STATISTICAL ANALYSIS PLAN

**Study Title:** A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety

and Efficacy of GS-9883/Emtricitabine/Tenofovir Alafenamide Versus Dolutegravir + Emtricitabine/Tenofovir Alafenamide in

HIV-1 Infected, Antiretroviral Treatment-Naïve Adults

Name of Test Drug: Bictegravir/Emtricitabine/Tenofovir Alafenamide

(B/F/TAF; GS-9883/F/TAF)

Study Number: GS-US-380-1490

**Protocol Version (Date):** Amendment 2 (21 October 2016)

**Analysis Type:** Week 48 Interim Analysis

**Analysis Plan Version:** Version 1.0

**Analysis Plan Date:** 10 May 2017

Analysis Plan Author(s): PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# **TABLE OF CONTENTS**

| TAB | LE OF | CONTENTS | 2 |
|---|---|---|---|
| LIST | OF IN | -TEXT TABLES | 4 |
| LIST | OF AE | BBREVIATIONS | 5 |
| PHA | RMAC | OKINETIC ABBREVIATIONS | 7 |
| 1. | INTRO | DDUCTION | 8 |
| | 1.1. | Study Objectives | 8 |
| | 1.2. | Study Design | |
| | 1.3. | Sample Size and Power | |
| 2. | TYPE | OF PLANNED ANALYSIS | |
| | 2.1. | Data Monitoring Committee Analyses | |
| | 2.2. | Interim Analyses | |
| | | 2.2.1. Week 46 Analysis | |
| | | 2.2.3. Week 144 Analysis | |
| | 2.3. | Final Analysis | |
| 3. | GENE | RAL CONSIDERATIONS FOR DATA ANALYSES | |
| ٥. | 3.1. | Analysis Sets | |
| | 3.1. | 3.1.1. All Randomized Analysis Set. | |
| | | 3.1.2. Full Analysis Set | |
| | | 3.1.3. Per Protocol Analysis Set | |
| | | 3.1.4. Safety Analysis Set | |
| | | 3.1.5. Pharmacokinetic Analysis Set | |
| | | 3.1.6. Pharmacokinetic Substudy Analysis Set | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates. | |
| | 3.4. | Examination of Subject Subgroups | |
| | | 3.4.1. Subject Subgroups for Efficacy Analyses | |
| | | 3.4.2. Subject Subgroups for Safety Analyses | |
| | 3.5. | Multiple Comparisons | |
| | 3.6. | Missing Data and Outliers | |
| | | 3.6.1. Missing Data | 16 |
| | | 3.6.2. Outliers | 16 |
| | 3.7. | Data Handling Conventions and Transformations | 16 |
| | 3.8. | Analysis Windows | 18 |
| | | 3.8.1. Definition of Study Day | 18 |
| | | 3.8.2. Analysis Windows | 18 |
| | | 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis | |
| | | Window | 21 |
| 4. | SUBJE | ECT DISPOSITION | 22 |
| | 4.1. | Subject Enrollment and Disposition | 22 |
| | | 4.1.1. Subject Enrollment | |
| | | 4.1.2. Subject Disposition | |
| | 4.2. | Extent of Study Drug Exposure and Adherence | |
| | | 4.2.1. Duration of Exposure to Study Drug | |
| | | 4.2.2. Adherence to Study Drug Regimen | |
| | 4.3. | Protocol Deviations | 24 |

| 5. | BASELINE CHARACTERISTICS | | |
|---|---|---|---|
| | 5.1. | Demographics and Baseline Characteristics | 25 |
| | 5.2. | Baseline Disease Characteristics | |
| | 5.3. | Medical History | |
| 6. | EFFIC | CACY ANALYSES | 27 |
| | 6.1. | Primary Efficacy Endpoint | 27 |
| | | 6.1.1. Definition of the Primary Efficacy Endpoint | |
| | | 6.1.2. US FDA-defined Snapshot Algorithm | |
| | | 6.1.3. Statistical Hypothesis for the Primary Efficacy Endpoint | |
| | | 6.1.4. Primary Analysis of the Primary Efficacy Endpoint | |
| | | 6.1.5. Secondary Analysis of the Primary Efficacy Endpoint | |
| | | 6.1.6. Subgroup Analysis of the Primary Efficacy Endpoint | |
| | 6.2. | Secondary Efficacy Endpoints | |
| | | 6.2.1. Definition of the Secondary Efficacy Endpoints | |
| | | 6.2.2. Analysis of the Secondary Efficacy Endpoints | |
| | 6.3. | Tertiary Efficacy Endpoints | |
| | | 6.3.1. Definition of the Tertiary Efficacy Endpoints | |
| | | 6.3.2. Analysis of the Tertiary Efficacy Endpoints | |
| | 6.4. | Changes From Protocol-Specified Efficacy Analyses | |
| 7. | SAFF | TTY ANALYSES | |
| | 7.1. | Adverse Events and Deaths | |
| | 7.1. | 7.1.1. Adverse Event Dictionary | |
| | | 7.1.2. Adverse Event Severity | |
| | | 7.1.3. Relationship of Adverse Events to Study Drug | |
| | | 7.1.4. Serious Adverse Events | |
| | | 7.1.5. Treatment-Emergent Adverse Events | |
| | | 7.1.6. Summaries of Adverse Events and Death | |
| | | 7.1.7. Additional Analysis of Adverse Events | |
| | 7.2. | Laboratory Evaluations | |
| | 1.2. | 7.2.1. Summaries of Numeric Laboratory Results | |
| | | 7.2.2. Graded Laboratory Values | |
| | | 7.2.3. Metabolic Laboratory Evaluations | |
| | | 7.2.4. Liver-Related Laboratory Evaluations | |
| | | 7.2.5. Renal-Related Laboratory Evaluations | |
| | 7.3. | Body Weight, Height, and Vital Signs | |
| | 7.4. | Prior and Concomitant Medications | |
| | / .¬. | 7.4.1. Nonstudy Drug Antiretroviral Medications | |
| | | 7.4.2. Concomitant Non-ARV Medications | |
| | 7.5. | Electrocardiogram Results | |
| | 7.6. | Other Safety Measures | |
| | 7.0.<br>7.7. | Changes From Protocol-Specified Safety Analyses | |
| 8. | | RMACOKINETIC ANALYSES | |
| | 8.1. Estimation of Pharmacokinetic Parameters | | |
| | 8.2. | Analysis for Intensive PK (PK Substudy Analysis Set) | |
| | 8.3. | Analysis for Trough and Postdose PK (PK Analysis Set) | |
| | 8.4. | Changes from Protocol-Specified Pharmacokinetic Analysis Set) | |
| 0 | | TAL POPULATION ANALYSES | |
| 9. | SPEC | | |
| | 9.1. | Analyses for HIV/HBV Coinfected Subjects | |
| | 9.2. | Analyses for HIV/HCV Coinfected Subjects | 48 |

| 10. | REFERENCES | | 49 |
|---|---|---|---|
| 11. | SOFTWARE | | 50 |
| 12. | SAP REVISION | V | 51 |
| 13. | APPENDICES | | 52 |
| | Appendix 1. | Study Procedures Table | 53 |
| | Appendix 2. | Flowchart of US FDA-defined Snapshot Algorithm (for Naïve Trial) | 58 |
| | Appendix 3. | Region Definition | 59 |
| | Appendix 4. | Selected Medical History | 60 |
| | Appendix 5. | Hepatic Events | 82 |
| | Appendix 6. | Programming Specification | 83 |
| | | LIST OF IN-TEXT TABLES | |
| | Table 3-1. | Subjects Excluded from Week 48 PP Analysis Set Due to Premature | |
| | | Discontinuation of Study Drug and/or Missing HIV-1 RNA Assessment in Week 48 | |
| | | Analysis Window | 13 |
| | Table 3-2. | Analysis Windows for HIV-1 RNA, CD4+ cell count, CD4 %, HBV DNA, | |
| | | Hematology, Chemistry, Urinalysis, and Urine Pregnancy Laboratory Tests, | • • |
| | m 11 0 0 | eGFR <sub>CG</sub> , Vital Signs, and Weight | |
| | Table 3-3. | Analysis Windows for Metabolic Assessments | |
| | Table 3-4. | Analysis Windows for TSH | |
| | Table 3-5. | Analysis Windows for HCV Serology and HCV RNA Assessments | |
| | Table 3-6. | Analysis Windows for Safety ECG | |
| | Table 8-1. | Treatment and Associated Analytes | 45 |

#### LIST OF ABBREVIATIONS

3TC lamivudine ABC abacavir

ABC/DTG/3TC fixed dose combination of abacavir (ABC) 600 mg / dolutegravir (DTG) 50 mg /

lamivudine (3TC) 300 mg

AE adverse event

ALP alkaline phosphatase
ALT alanine aminotransferase
ANOVA analysis of variance

ARV antiretroviral

ART antiretroviral treatment
AST aspartate aminotransferase

BIC bictegravir

B/F/TAF fixed dose combination of bictegravir (BIC; B) 50 mg / emtricitabine (FTC; F) 200 mg /

tenofovir alafenamide (TAF) 25 mg

BLQ below limit of quantitation

BMI body mass index

CDER Center for Drug Evaluation and Research

CG Cockcroft-Gault
CI confidence interval

CMH Cochran-Mantel-Haenszel

CRF case report form
CSR clinical study report
CV coefficient of variation

DC premature study drug discontinuation

DNA deoxyribonucleic acid

DSPH Drug Safety and Public Health

DTG dolutegravir, tivicay ECG electrocardiogram

eCRF electronic case report form

eGFR estimated glomerular filtration rate

eGFR<sub>CG</sub> estimated glomerular filtration rate using Cockcroft-Gault formula

FAS full analysis set

FDA Food and Drug Administration

FDC fixed dose combination

F/TAF fixed dose combination of emtricitabine (FTC; F)/ tenofovir alafenamide (TAF)

FTC, F emtricitabine

GEN Genvoya, E/C/F/TAF
GFR glomerular filtration rate
Gilead Gilead Sciences, Inc.

GS-9883 bictegravir

HBcAb hepatitis B core antibody
HBeAb hepatitis B e-antibody
HBeAg hepatitis B e-antigen

HBsAb hepatitis B surface antibody HBsAg hepatitis B surface antigen

HBV hepatitis B virus
HCV hepatitis C virus
HCVAb hepatitis C antibody
HDL high density lipoprotein

HIV-1 human immunodeficiency virus (Type 1)

HLGT high level group term HLT high level term

ICH International Conference on Harmonisation of Technical Requirements for Registration of

Pharmaceuticals for Human Use

ID identification

IDMC independent data monitoring committee

IWRS interactive web response system

LDL low density lipoprotein LLT lowest level term

MedDRA Medical Dictionary for Regulatory Activities

MH Mantel-Haenszel

PEP post-exposure prophylaxis
PrEP pre-exposure prophylaxis

PK pharmacokinetic
PP per protocol
PT preferred term
Q quartile

Q1 first quartile
Q3 third quartile
QD once daily
RNA ribonucleic acid
SAE serious adverse events
SAP statistical analysis plan

SMQ Standardised MedDRA Query

SOC system organ class
TAF tenofovir alafenamide
TFL tables, figures, and listings

TFV tenofovir

SD

TSH thyroid stimulating hormone; thyrotropin

standard deviation

ULN upper limit of normal WHO World Health Organization

#### PHARMACOKINETIC ABBREVIATIONS

AUC<sub>last</sub> area under the concentration versus time curve from time zero to the last quantifiable

concentration

AUC<sub>tau</sub> area under the concentration versus time curve over the dosing interval

C<sub>last</sub> last observed quantifiable concentration of the drug in plasma

C<sub>max</sub> maximum observed concentration of drug in plasma

C<sub>tau</sub> observed drug concentration at the end of the dosing interval CLss/F apparent oral clearance after administration of the drug:

at steady state:  $CLss/F = Dose/AUC_{tau}$ , where "Dose" is the dose of the drug

LAMBDAZ ( $\lambda_z$ ) terminal elimination rate constant, estimated by linear regression of the terminal elimination

phase of the plasma concentration of drug versus time curve

THALF (t<sub>1/2</sub>) estimate of the terminal elimination half-life of the drug in plasma, calculated by dividing

the natural log of 2 by the terminal elimination rate constant  $(\lambda_z)$ 

 $T_{last}$  time (observed time point) of  $C_{last}$   $T_{max}$  time (observed time point) of  $C_{max}$ 

V<sub>z</sub>/F apparent volume of distribution of the drug

### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) of the Week 48 interim analysis for Study GS-US-380-1490, which will be performed when all subjects have completed their Week 48 visit or prematurely discontinued from the study drug. This SAP is based on the study protocol amendment 2 dated 21 October 2016 and the electronic case report form (eCRF). The SAP will be finalized before database finalization for the interim analysis. Any changes made after the finalization of the SAP will be documented in the clinical study report (CSR).

# 1.1. Study Objectives

The primary objective of this study is:

• To evaluate the efficacy of a fixed dose combination (FDC) containing bictegravir (GS-9883; BIC; B) /emtricitabine (FTC; F) /tenofovir alafenamide (TAF) versus dolutegravir (DTG) + a FDC containing emtricitabine/tenofovir alafenamide (F/TAF) in HIV-infected, antiretroviral treatment (ART)-naïve adult subjects as determined by the achievement of HIV-1 ribonucleic acid (RNA) < 50 copies/mL at Week 48.

The secondary objectives of this study are:

• To evaluate the efficacy, safety, and tolerability of the 2 treatment groups through Weeks 48, 96, and 144.

### 1.2. Study Design

#### **Design Configuration and Subject Population**

GS-US-380-1490 is a randomized, double-blinded, multicenter, active-controlled study to evaluate the safety and efficacy of B/F/TAF FDC versus DTG + F/TAF FDC in HIV-infected ART-naive adult subjects.

#### **Treatment Groups**

Subjects who provide written consent and meet all eligibility criteria will be randomized in a 1:1 ratio to one of the following 2 treatment groups:

- **Treatment Group 1:** FDC of bictegravir 50 mg/ emtricitabine 200 mg/ tenofovir alafenamide 25 mg (B/F/TAF) + Placebo to match dolutegravir 50 mg and Placebo to match FDC of emtricitabine 200 mg/tenofovir alafenamide 25 mg (F/TAF) administered orally, once daily, without regard to food (n = 300)
- **Treatment Group 2:** Dolutegravir 50 mg + FDC of emtricitabine 200 mg/tenofovir alafenamide 25 mg (F/TAF) + Placebo to match FDC of bictegravir 50 mg/ emtricitabine 200 mg/ tenofovir alafenamide 25 mg (B/F/TAF) administered orally, once daily, without regard to food (n = 300)

# **Key Eligibility Criteria**

Medically stable HIV-infected subjects who meet the following criteria:

- Plasma HIV-1 RNA levels  $\geq$  500 copies/mL at screening
- ART-naive (≤ 10 days of prior therapy with any antiretroviral [ARV] agent following a diagnosis of HIV-1 infection) except the use for pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP), up to 1 month prior to screening.
- Screening genotype report must show sensitivity to FTC and tenofovir (TFV)
- Estimated GFR ≥ 30 mL/min according to the Cockcroft-Gault formula for creatinine clearance

#### **Study Periods / Phases**

Subjects will be treated for at least 144 weeks during the blinded treatment phase. After Week 144, all subjects will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Once the last subject completes the Week 144 visit and Gilead Sciences Inc. (Gilead) completes the Week 144 analysis, all subjects will return to the clinic (preferably within 30 days) for an End of Blinded Treatment Visit. At the End of Blinded Treatment Visit, if safety and efficacy of B/F/TAF FDC are demonstrated following review of unblinded data, subjects in a country where B/F/TAF FDC is not available will be given the option to receive B/F/TAF FDC in an open label (OL) extension phase for up to 48 weeks, or until the product becomes accessible to subjects through an access program, or until Gilead elects to discontinue the study in that country, whichever occurs first.

All subjects participating in the OL extension phase, without regard to their blinded treatment regimen, will return for study visits at Week 12 OL and every 12 weeks thereafter for up to 48 weeks.

Subjects who complete the study through the End of Blinded Treatment Visit and do not continue on the OL B/F/TAF FDC extension phase will be required to return to the clinic after the End of Blinded Treatment Visit for a 30-Day Follow-Up Visit.

Treatment assignments will be provided to the investigators within 30 days of the last subject completing the End of Blinded Treatment Visit.

### **Schedule of Assessments**

After screening procedures, eligible subjects will be randomized 1:1 to Treatment Group 1 or Treatment Group 2 and treated for 144 weeks. Following the Day 1 visit, subjects will be required to return for study visits at Weeks 4, 8, and 12, and then every 12 weeks from Week 12 through Week 144. After Week 144, all subjects will continue to take their blinded study drugs and attend study visits every 12 weeks until the End of Blinded Treatment Visit.

For all eligible subjects, blood will be collected at Day 1, Weeks 4, 8, 12, and then every 12 weeks through the End of Blinded Treatment Visit. Laboratory analyses (hematology, chemistry, and urinalysis), HIV-1 RNA, CD4+ cell count, and complete or symptom directed physical examinations will be performed at Screening, Day 1 and all subsequent visits.

Adverse events and concomitant medications will be assessed at each visit.

More details for study procedures could be found in Appendix 1.

#### **Pharmacokinetics**

An intensive pharmacokinetic (PK) substudy will be performed at the Week 4 or 8 visit in a subset of subjects (target n = 30) at study sites able to conduct this testing.

For all subjects on study drug, a single anytime pre- or post-dose PK blood sample will be collected at Weeks 8, 24, and 36.

For all subjects on study drug, a trough PK blood sample will be obtained 20-28 hours following the last dose at Weeks 4 and 12. Following an observed dose, one post-dose PK blood sample will be collected between 1 and 4 hours post-dose.

## **Randomization**

Subjects will be randomized in a 1:1 ratio to 1 of 2 Treatment Groups (Treatment Group 1: Treatment Group 2). Randomization will be stratified by HIV-1 RNA level (\$\leq\$ 100,000 copies/mL, \$\rightarrow\$ 100,000 to \$\leq\$ 400,000 copies/mL, or \$\rightarrow\$ 400,000 copies/mL) at screening, CD4+ cell count (\$\leq\$ 50 cells/\muL, 50 - 199 cells/\muL, or \$\geq\$ 200 cells/\muL) at screening, and region (US or Ex-US) at randomization.

### **Site and/or Stratum Enrollment Limits**

Approximately 150 study sites in North America, Europe, and Latin America participated. There was no enrollment limit for individual sites.

# Study Duration

The randomized, double-blind phase of this study is at least 144 weeks in duration.

### 1.3. Sample Size and Power

A total of approximately 600 HIV-infected subjects, randomized in a 1:1 ratio to 2 treatment groups (300 subjects per treatment group), achieves at least 95% power to detect a noninferiority margin of 12% in Week 48 response rate (HIV-1 RNA < 50 copies/mL as determined by the United States [US] Food and Drug Administration [FDA]-defined snapshot algorithm) difference between the 2 treatment groups. For sample size and power computation, it is assumed that both treatment groups have a response rate of 91% (based on Gilead Genvoya [GEN; E/C/F/TAF] Studies GS-US-292-0104 and GS-US-292-0111), that a noninferiority margin is 12%, and that the significance level of the test is at a one-sided 0.025 level. Sample size and power calculations were made using the statistical software package nQuery Advisor (Version 6.0).

### 2. TYPE OF PLANNED ANALYSIS

# **2.1.** Data Monitoring Committee Analyses

The Week 12 Independent Data Monitoring Committee (IDMC) analysis was conducted after approximately the first 50% of subjects enrolled completed their Week 12 visit or prematurely discontinued the study drug. The Week 24 IDMC analysis was conducted after all subjects enrolled completed their Week 24 visit or prematurely discontinued the study drug. The purpose of these interim analyses was to provide the IDMC with a statistical report for review. More details are documented in the IDMC charter.

Gilead does not have a prior intent to ask the IDMC to review Week 48 results or to consider early termination of the study even if there is early evidence of favorable efficacy for B/F/TAF.

### 2.2. Interim Analyses

# 2.2.1. Week 48 Analysis

The Week 48 analysis will be conducted after all subjects either complete their Week 48 visit or prematurely discontinue from the study drug.

This statistical analysis plan describes the analysis plan for the Week 48 interim analysis, the primary analysis of this study.

#### 2.2.2. Week 96 Analysis

The Week 96 analysis will be conducted after all subjects either complete their Week 96 visit or prematurely discontinue from the study drug.

## 2.2.3. Week 144 Analysis

The Week 144 analysis will be conducted after all subjects either complete their Week 144 visit or prematurely discontinue from the study drug.

## 2.3. Final Analysis

The final statistical analysis will be conducted after all subjects either complete the study or prematurely discontinue from the study.

### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (SD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

All statistical tests will be 2-sided and performed at the 5% significance level unless otherwise specified.

By-subject listings will be presented for all subjects in the All Randomized analysis set unless otherwise specified, and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as AEs, will be presented in chronological order within a subject. The treatment group to which subjects were randomized will be used in the listings.

In general, age (in years) on the date of the first dose of study drug will be used for analyses and presentation in listings. For randomized but never dosed subjects, age on the date of randomization will be used. For screen failures, age on the date of the informed consent was signed will be used. If only birth year is collected on the eCRF, "01 January" will be used for the unknown birth day and month for the purpose of age calculation, similarly, if only birth year and month are collected on the eCRF, "01" will be used for the unknown birth day for the purpose of age calculation.

In general, permanent discontinuation of study drug refers to premature discontinuation of study drug or completion of study drug.

#### 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. Subjects included in each analysis set will be determined before the study blind is broken for analysis. The analysis set will be included as a subtitle of each table, figure, and listing. A summary of the number and percentage of subjects in each analysis set will be provided by treatment group and in total.

#### 3.1.1. All Randomized Analysis Set

The **All Randomized Analysis Set** will include all subjects who are randomized into the study. This is the primary analysis set for by-subject listings.

#### 3.1.2. Full Analysis Set

The **Full Analysis Set (FAS)** will include all subjects who (1) are randomized into the study and (2) have received at least 1 dose of study drug. Subjects will be grouped according to the treatment to which they were randomized. For the FAS, all efficacy data, including data collected after the last dose of study drug, will be included, unless specified otherwise. This is the primary analysis set for efficacy analyses.

# 3.1.3. Per Protocol Analysis Set

The Week 48 **Per Protocol (PP) Analysis Set** will include all subjects who (1) are randomized into the study, (2) have received at least 1 dose of study drug, and (3) have not committed any major protocol violation, including the violation of key entry criteria. Subjects will be grouped according to the treatment they actually received. For the PP analysis, efficacy data up to 1 day after permanent discontinuation of study drug will be included. The Week 48 PP analysis set is the secondary analysis set for efficacy analysis.

Subjects meeting any of the following criteria will be excluded from the Week 48 PP analysis set:

• Subjects who do not have on-treatment HIV-1 RNA in the Week 48 analysis window, except when missing is due to discontinuation of study drug for lack of efficacy. (Note: lack of efficacy is defined as having the check-box for Lack of Efficacy marked as the reason for premature study drug discontinuation in the "Blinded Treatment" study phase on the study drug completion eCRF page; Table 3-1).

Table 3-1. Subjects Excluded from Week 48 PP Analysis Set Due to Premature Discontinuation of Study Drug and/or Missing HIV-1 RNA Assessment in Week 48 Analysis Window

| Discontinuation from Stud | dy Drug prior to or on the | HIV-1 RNA Data on Randomized Treatment<br>Available in Week 48 Analysis Window | |
|---|---|---|---|
| Upper Bound of Week 48 Analysis Window | | Yes | No |
| Yes | Due to Lack of Efficacy | + | + |
| res | Due to Other Reasons | + | <del>-</del> |
| No | | + | <del>-</del> |

<sup>+=</sup> Inclusion of Subjects in Week 48 PP analysis set; -= Exclusion of Subjects in Week 48 PP analysis set.

- Subjects who do not meet the inclusion criterion that the screening genotype report must show sensitivity to FTC and, TFV
- Subjects who meet the exclusion criterion for receiving ongoing therapy with any of the medications listed in the table in protocol Section 4.3 including drugs not to be used with BIC, FTC, TAF, and DTG
- Nonadherence to study drug: subjects with adherence rate for active study drug up to the Week 48 Visit below the 2.5th percentile

#### 3.1.4. Safety Analysis Set

The **Safety Analysis Set** will include all subjects who (1) are randomized into the study and (2) have received at least 1 dose of study drug. All the data collected up to 30 days after permanent discontinuation of the study drug will be included in the safety summaries, unless specified otherwise. Subjects will be grouped according to the treatment they actually received. This is the primary analysis set for safety analyses.

# 3.1.5. Pharmacokinetic Analysis Set

The **PK** Analysis Set will include all subjects who (1) are randomized into the study, (2) have received at least 1 dose of active B/F/TAF, and (3) have at least 1 nonmissing PK concentration value for any analyte of interest reported by the PK lab. The PK analysis set will be used for general PK analyses.

# 3.1.6. Pharmacokinetic Substudy Analysis Set

The **PK** Substudy Analysis Set will include all subjects who (1) are randomized into the study, (2) are enrolled into the PK Substudy, (3) have received at least 1 dose of active B/F/TAF, and (4) have at least 1 nonmissing intensive PK concentration value for any analyte of interest reported by the PK lab. The PK substudy analysis set will be used for intensive PK analyses.

## 3.2. Subject Grouping

For analyses based on the All Randomized Analysis Set or the FAS, subjects will be grouped by randomized treatment. For other analyses, subjects will be grouped by actual treatment received. The actual treatment received will differ from the randomized treatment only when the actual treatment received differs from randomized treatment for the entire treatment duration.

#### 3.3. Strata and Covariates

Randomization was stratified by HIV-1 RNA level ( $\leq 100,000$  copies/mL, > 100,000 copies/mL to  $\leq 400,000$  copies/mL, or > 400,000 copies/mL) at screening, CD4+ cell count (< 50 cells/ $\mu$ L, 50 - 199 cells/ $\mu$ L, or  $\geq 200$  cells/ $\mu$ L) at screening, and region (US or Ex-US) at randomization.

Efficacy analyses will include 2-level HIV-1 RNA stratum ( $\leq$  100,000 vs. > 100,000 copies/mL) at baseline and region stratum (US vs. Ex-US) at randomization as stratification factors. The CD4+ cell count stratum was excluded for the analysis due to the following reasons: (1) HIV-1 RNA level and CD4+ cell count are highly correlated; (2) a balanced CD4+ cell count distribution between treatment groups is expected since CD4+ cell count was one of the stratification factors used during the randomization; and (3) the risk of including small or missing stratum during the analysis will be reduced. The HIV-1 RNA stratum will be reclassified using baseline HIV-1 RNA level for analysis purposes. Furthermore, since the number of subjects in the HIV-1 RNA > 400,000 copies/mL stratum is small, this stratum will be combined with HIV-1 RNA > 100,000 to  $\leq$  400,000 copies/mL stratum to form a 2-level HIV-1 RNA stratum ( $\leq$  100,000 vs. > 100,000 copies/mL). This will prevent small or missing stratum during the analysis.

## 3.4. Examination of Subject Subgroups

## 3.4.1. Subject Subgroups for Efficacy Analyses

The proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 determined by the US FDA-defined snapshot algorithm {U. S. Department of Health and Human Services 2015} will be analyzed for the following subject subgroups (see Section 6.1.6 for details):

- Age (years): (a) < 50 and (b)  $\ge 50$
- Sex: (a) male and (b) female
- Race: (a) black and (b) nonblack
- Baseline HIV-1 RNA level (copies/mL): (a)  $\leq 100,000$  and (b) > 100,000
- Baseline CD4+ cell count (/ $\mu$ L): (a) < 200 and (b)  $\geq$  200
- Region: (a) US and (b) Ex-US
- Study drug adherence (%): (a)  $\leq$  95 and (b)  $\geq$  95 (based on adherence up to Week 48 visit)

The proportion of subjects with HBV Deoxyribonucleic Acid (DNA) < 29 IU/mL at baseline and Week 48, and the change from baseline in log10 HBV DNA by visit will be analyzed for the following subject subgroup:

• Subjects with HIV/HBV coinfection at baseline

## 3.4.2. Subject Subgroups for Safety Analyses

Selected safety endpoints may be analyzed for the following subject subgroups (see Section 9.1 for details):

- Subjects with HIV/HBV coinfection at baseline
- Subjects with incident HIV/HBV coinfection while on study drug (if any)

Selected safety endpoints will be analyzed for the following subject subgroups (see Section 9.2 for details):

- Subjects with HIV/hepatitis C virus (HCV) coinfection at baseline
- Subjects with incident HIV/HCV coinfection while on study drug (if any)

#### 3.5. **Multiple Comparisons**

The noninferiority evaluation of the proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm was the prespecified primary comparison. However, 2 interim IDMC analyses were performed prior to the analysis for the primary endpoint and an alpha penalty of 0.00001 was applied for each interim IDMC meeting. Therefore, the alpha level for the primary endpoint (ie, the proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm) was adjusted to 0.04998 (corresponding to 95.002% confidence interval [CI]) using both the FAS and the Week 48 PP analysis set. No alpha level adjustment is applied other than for the primary endpoint.

#### 3.6. **Missing Data and Outliers**

#### 3.6.1. **Missing Data**

A missing datum for a given study analysis window may be due to any of the following reasons:

- A visit occurring in the window but data were not collected or were unusable
- A visit not occurring in the window
- A subject prematurely discontinuing from the study before reaching the window

In general, values for missing data will not be imputed, unless methods for handling missing data are specified.

For missing last dosing date of study drug, imputation rules are described in Section 3.8.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.5.2, and for concomitant medications in Section 7.4.1.

#### 3.6.2. **Outliers**

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be done to evaluate the impact of outliers on efficacy or safety outcomes, unless specified otherwise. All data will be included in the analyses.

#### 3.7. **Data Handling Conventions and Transformations**

Laboratory data that are continuous in nature but are less than the lower limit of quantitation or above the upper limit of quantitation will be imputed as follows except for urine creatinine:

A value that is 1 unit less than the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (where x is considered the limit of quantitation). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used for calculation of summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used for calculation of summary statistics.

- A value that is 1 unit above the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (where x is considered the limit of quantitation). Values with decimal points will follow the same logic as above.
- The limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the limit of quantitation).

Logarithmic (base 10) transformations will be applied to HIV-1 RNA and HBV DNA data for efficacy analyses. HIV-1 RNA results of 'No HIV-1 RNA detected' and "<20 cp/mL HIV-1 RNA Detected" will be imputed as 19 copies/mL for analysis purposes. HBV DNA results of "<20 IU/mL HBV DNA detected" or "No HBV DNA detected" will be imputed as 19 IU/mL for analysis purposes. HCV RNA results of "<15 IU/mL HCV RNA detected" or "No HCV RNA detected" will be imputed as 14 IU/mL for analysis purposes.

Natural logarithmic transformations will be used for analyzing concentrations and PK parameters in intensive plasma samples. Concentration values (including intensive, trough, predose, postdose, anytime PK concentration) that are below the lower limit of quantitation (BLQ) will be presented as "BLQ" in the concentration listing. Intensive PK concentration values that are BLQ will be treated as 0 at predose time points and one-half the value of the lower limit of quantitation (LLOQ) at postdose time points for summary purposes. Other PK concentration values (including trough, predose, postdose, anytime PK concentration) that are BLQ will be treated as one-half of the LLOQ.

The following conventions will be used for the presentation of order statistics and summary statistics for intensive PK concentration:

- If at least 1 subject has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the subjects have a concentration value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."
- If more than 50% of the subjects have a concentration value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the subjects have a concentration value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all subjects have concentration values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) and summary statistics will be displayed as "BLQ."

# 3.8. Analysis Windows

## 3.8.1. Definition of Study Day

**Study Day 1** is defined as the day when the first dose of study drug (ie, B/F/TAF or Placebo, DTG + F/TAF or Placebo) was taken, as recorded on the Study Drug Administration eCRF form.

**Study Days** are calculated relative to Study Day 1. For events that occurred on or after the Study Day 1 date, study days are calculated as (visit date minus Study Day 1 plus 1). For events that occurred prior to Study Day 1, study days are calculated as (visit date minus Study Day 1).

**Last Dose Date** is the latest of the blinded study drug end dates recorded on the Study Drug Administration eCRF form with "Permanently Withdrawn" box checked for subjects who prematurely discontinued or completed study drug in the "Blinded Treatment" study phase according to the Study Drug Completion eCRF.

If last dose date is missing (eg, only year of last dose date is known or completely missing due to lost to follow-up) for subjects who prematurely discontinued or completed blinded study drug at the data cut date, the latest of the study drug start dates and end dates, the clinical visit dates, and the laboratory visit dates, excluding the date of 30-day follow-up visit, will be used to impute the last dose date. For other partial missing last dose date, please see the programming specifications for imputation rule details.

**Last Study Date** is the latest of the study drug start dates and end dates, the clinic visit dates, and the laboratory visit dates, including the 30-day follow-up visit date, for subjects who prematurely discontinued study or who completed study according to the Study Completion eCRF.

**Baseline value** is defined as the last value obtained on or prior to Study Day 1 for all assessments.

# 3.8.2. Analysis Windows

Subject visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

The analysis windows for HIV-1 RNA, CD4+ cell count, CD4 %, HBV DNA, hematology, chemistry, urinalysis, urine pregnancy laboratory tests, eGFR<sub>CG</sub>, vital signs, and weight are presented in Table 3-2. Note: HBV DNA is only collected at Baseline, Week 48, and every 48 weeks for subjects who are not HBV infected at any visit.

Table 3-2. Analysis Windows for HIV-1 RNA, CD4+ cell count, CD4 %, HBV DNA, Hematology, Chemistry, Urinalysis, and Urine Pregnancy Laboratory Tests, eGFR<sub>CG</sub>, Vital Signs, and Weight

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline | | | 1 |
| Week 4 | 28 | 2 | 42 |
| Week 8 | 56 | 43 | 70 |
| Week 12 | 84 | 71 | 126 |
| Week 24 | 168 | 127 | 210 |
| Week 36 | 252 | 211 | 294 |
| Week 48 | 336 | 295 | 378 |
| Week 60 | 420 | 379 | 462 |
| Week 72 | 504 | 463 | 546 |
| Week 84 | 588 | 547 | 630 |
| Week 96 | 672 | 631 | 714 |
| Week 108 | 756 | 715 | 798 |
| Week 120 | 840 | 799 | 882 |
| Week K (K is every 12 weeks after previous visit) | K*7 | (K-6)*7+1 | (K+6)*7 |

The analysis windows for metabolic assessments (including fasting glucose and lipid panel: total cholesterol, high density lipoprotein [HDL], direct low density lipoprotein [LDL], triglycerides, and total cholesterol to HDL ratio) and HBV serology (including hepatitis B surface antibody [HBsAb], hepatitis B surface antigen [HBsAg], hepatitis B e-antigen [HBeAg], and reflex hepatitis B e-antibody [HBeAb] if HBeAg is negative, for subjects who are HBV infected at any visit and HBsAb, HBcAb, HBsAg, for those subjects who do not meet the definition of HBV infection at any visit) are presented in Table 3-3. Note: HBV serology is only collected at Baseline, Week 48, and every 48 weeks for subjects who are not HBV infected at any visit.

Table 3-3. Analysis Windows for Metabolic Assessments

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline | | | 1 |
| Week 12 | 84 | 2 | 126 |
| Week 24 | 168 | 127 | 252 |
| Week 48 | 336 | 253 | 420 |
| Week 72 | 504 | 421 | 588 |
| Week 96 | 672 | 589 | 756 |
| Week 120 | 840 | 757 | 924 |
| Week K (K is every 24 weeks after previous visit) | K*7 | (K-12)*7+1 | (K+12)*7 |

The analysis windows for thyroid stimulating hormone (TSH; thyrotropin) is presented in Table 3-4.

Table 3-4. Analysis Windows for TSH

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline | | | 1 |
| Week 24 | 168 | 2 | 252 |
| Week 48 | 336 | 253 | 420 |
| Week 72 | 504 | 421 | 588 |
| Week 96 | 672 | 589 | 756 |
| Week 120 | 840 | 757 | 924 |
| Week 144 | 1008 | 925 | 1092 |
| Week K (K is every 24 weeks after previous visit) | K*7 | (K-12)*7+1 | (K+12)*7 |

The analysis windows for HCV serology (HCV antibody [HCVAb]) and HCV RNA assessments are presented in Table 3-5.

Table 3-5. Analysis Windows for HCV Serology and HCV RNA Assessments

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline | | | 1 |
| Week 48 | 336 | 2 | 504 |
| Week 96 | 672 | 505 | 840 |
| Week K (K is every 48 weeks after previous visit) | K*7 | (K-24)*7+1 | (K+24)*7 |

The analysis windows for safety electrocardiogram (ECG) are presented in Table 3-6.

Table 3-6. Analysis Windows for Safety ECG

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline | | | 1 |
| Week 24 | 168 | 2 | 252 |
| Week 48 | 336 | 253 | 504 |
| Week 96 | 672 | 505 | 840 |
| Week K (K is every 48 weeks after previous visit) | K*7 | (K-24)*7+1 | (K+24)*7 |

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Window

Depending on the statistical analysis method, single values are required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time to event analysis would not require one value per analysis window. When a single value is needed, the following rule(s) will be used.

If multiple nonmissing numeric observations exist in a window, then records will be chosen as follows:

- For baseline, the latest available record on or prior to the first dose date of study drug will be selected. If there are multiple records with the same time or no time recorded on the same day, average will be used for the baseline value, except for HIV-1 RNA (see below).
- For postbaseline visits:
  - For CD4+ cell count, CD4%, HBV DNA, the record(s) collected on the latest day in the window will be selected for analysis.
  - For other numeric observations (ie, except HIV-1 RNA, CD4+ cell count, CD4%, and HBV DNA), the record(s) collected on the day closest to the nominal day for that visit will be selected. If there are 2 days equidistant from the nominal day, the later day will be selected.
  - For any numeric observations except HIV-1 RNA, if there are multiple records on the selected day, the average will be taken.
- For baseline and postbaseline HIV-1 RNA, the latest (considering both date and time) record(s) in the window will be selected. If both "HIV RNA Taqman 2.0" and "HIV RNA Repeat" (ie, the HIV-1 RNA result obtained from an additional aliquot of the original sample) are available with the same collection time, the results from the "HIV RNA Repeat" will be selected for analysis purposes; otherwise, if there are multiple "HIV RNA Taqman 2.0" records with the same collection time, the geometric mean will be taken for analysis purposes.

If multiple valid nonmissing categorical observations exist in a window, records will be chosen as follows:

- For baseline, the last available record on or prior to the first dose date of study drug will be selected. If there are multiple records with the same time or no time recorded on the same day, the value with the lowest severity will be selected (eg, normal will be selected over abnormal for safety ECG findings).
- For postbaseline visits, the most conservative value within the window will be selected (eg, abnormal will be selected over normal for safety ECG findings).

## 4. SUBJECT DISPOSITION

# 4.1. Subject Enrollment and Disposition

### 4.1.1. Subject Enrollment

The number and percentage of subjects randomized at each region, country, and investigator will be summarized by treatment group and overall using the safety analysis set. The region definition is provided in Appendix 3. The denominator for this calculation will be the number of subjects in the safety analysis set. Similarly, the number and percentage of subjects enrolled in each randomization stratum will be summarized based on reclassified strata using screening HIV-1 RNA and CD4+ Cell Count data instead of using interactive web response system (IWRS) data.

If there are discrepancies between IWRS and laboratory data with regard to stratum assignment, a listing of the discrepancies will be provided. If there are differences between randomization stratum using screening HIV-1 RNA value and baseline HIV-1 RNA value, a listing of the differences will be provided.

#### 4.1.2. Subject Disposition

The summary of subject disposition will be provided by treatment group and overall for all screened subjects. This summary will include the number of subjects screened, screen failure subjects who were not randomized, subjects who met all eligibility criteria and were not randomized, subjects randomized but never treated, subjects in the safety analysis set, and subjects in the FAS.

In addition, the number and percentage of the subjects in the following categories will be summarized:

- Still on study drug up to the data cut date
- Prematurely discontinuing study drug prior to the data cut date (with summary of reasons for discontinuing study drug)
- Still on study up to the data cut date
- Prematurely discontinuing from study prior to the data cut date (with summary of reasons for discontinuing study).

The denominator for the percentages of subjects in each category will be the number of subjects in the safety analysis set.

No inferential statistics will be generated. A data listing of reasons for premature study drug/study discontinuation will be provided.

# 4.2. Extent of Study Drug Exposure and Adherence

# 4.2.1. Duration of Exposure to Study Drug

Duration of exposure to study drug will be defined as (the last dose date – the first dose date + 1), regardless of temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks). For the calculation of the duration of exposure to study drug, the data cut date will be used to impute the last dose date for subjects who have not permanently discontinued study drug at the time of the data cut date.

Duration of exposure to study drug will be summarized using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) and as the number and percentage of subjects exposed for specified periods, eg,  $\geq$  4 weeks (28 days),  $\geq$  8 weeks (56 days),  $\geq$  12 weeks (84 days),  $\geq$  24 weeks (168 days),  $\geq$  36 weeks (252 days),  $\geq$  48 weeks (336 days),  $\geq$  60 weeks (420 days),  $\geq$  72 weeks (504 days),  $\geq$  84 weeks (588 days),  $\geq$  96 weeks (672 days),  $\geq$  108 weeks (756 days),  $\geq$  120 weeks (840 days),  $\geq$  132 weeks (924 days),  $\geq$  144 weeks (1008 days), etc.

Summaries will be provided by treatment group for subjects in the safety analysis set. No inferential statistics will be provided.

Time to permanent discontinuation of study drug will be analyzed using the Kaplan-Meier method by treatment group based on the safety analysis set. The log rank test will be used to compare the difference in study drug exposure between the 2 treatment groups. Subjects who are still on the randomized study drug will be censored on the imputed last dose date as defined in this section. A plot of KM estimates for the time to premature discontinuation of study drug by treatment group will be generated.

# 4.2.2. Adherence to Study Drug Regimen

Study drug regimen adherence will be computed based on pill counts for active drug only (eg, study drug regimen in Treatment Group 1 includes 1 study drug: B/F/TAF active. Study drug regimen in Treatment Group 2 includes 2 study drugs: DTG active + F/TAF active). The numbers of pills of study drug dispensed and returned are captured on study drug accountability eCRF.

Adherence (%) of study drug regimen will be calculated as follows:

Adherence (%) = 
$$100 \times \frac{\text{Total No. of pills taken}}{\text{Total No. of pills prescribed}}$$
  
=  $100 \times \frac{\sum \sum \text{No. of pills taken at each dispensing period}^{[1]}}{\sum \sum \text{No. of pills prescribed at each dispensing period}^{[2]}}$ 

- [1] Number of pills taken at a distinct dispensing period for a study drug is calculated as the minimum of (a) the daily number of pills prescribed for the study drug multiplied by the duration of treatment at the dispensing period, and (b) the number of pills taken for the study drug (number of pills dispensed minus the number of pills returned). Total number of pills taken is determined by summing the number of pills taken for each study drug contained in the study drug regimen from all evaluable dispensing periods.
- [2] Number of pills prescribed at a distinct dispensing period for a study drug is calculated as the daily number of pills prescribed for the study drug multiplied by the duration of treatment at the dispensing period. Total number of pills prescribed is determined by summing the number of pills prescribed for each study drug contained in the study drug regimen from all evaluable dispensing periods.

The duration of treatment at a dispensing period for a study drug is calculated as the minimum of (a) the last returned date of study drug at a dispensing period, (b) date of premature discontinuation of the study drug, and (c) <u>next pill dispensing date</u> of the study drug, minus dispensing date of the study drug.

The next pill dispensing date is the following dispensing date of the study drug regardless of the bottle return date.

For a record where the number of pills returned was missing (with "Yes" answered for "Was Bottle returned?" question), it is assumed the number of pills returned was zero. If the number of pills dispensed was missing or any study drug bottle was not returned or the bottle return status was unknown, then all records in that dispensing period for that study drug will be excluded from both denominator and numerator calculation.

Adherence up to the data cut date will be calculated using all data from the entire dosing period up to the date of permanent discontinuation of the study drug for subjects who prematurely discontinued study drug or completed study drug, or using all data available for subjects who are ongoing on study drug.

Adherence up to Week 48 visit will also be calculated using all data from the entire dosing period up to the date of permanent discontinuation of the study drug for subjects who prematurely discontinued study drug or completed study drug, or the Week 48 study drug dispensing date, whichever occurs earliest.

Descriptive statistics for adherence up to the data cut date and adherence up to Week 48 visit for a study drug regimen (n, mean, SD, median, Q1, Q3, minimum, and maximum) along with the number and percentage of subjects belonging to adherence categories (eg, < 80%,  $\ge 80\%$  to < 90%,  $\ge 90\%$  to < 95%,  $\ge 95\%$ ) will be provided by treatment group for subjects who return at least 1 bottle and have calculable adherence during the study in the safety analysis set. No inferential statistics will be provided.

#### 4.3. Protocol Deviations

A listing will be provided for all randomized subjects who violated at least 1 inclusion or exclusion criterion. The listing will include the criteria not met. A listing of subjects who received the wrong study drug will also be provided.

## 5. BASELINE CHARACTERISTICS

# 5.1. Demographics and Baseline Characteristics

Subject demographic data (eg, age, sex at birth, race, and ethnicity) and baseline characteristics (eg, body weight, height, and body mass index [BMI]) will be summarized by treatment group and overall using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) for continuous data and by the number and percentage of subjects for categorical data. The summaries of demographic data and baseline subject characteristics will be provided for the safety analysis set.

For categorical data, the Cochran-Mantel-Haenszel (CMH) test (ie, general association statistic for nominal data) will be used to compare the 2 treatment groups. For continuous data, the 2-sided Wilcoxon rank sum test will be used to compare the 2 treatment groups.

#### **5.2.** Baseline Disease Characteristics

The following baseline disease characteristics will be summarized by treatment group and overall using descriptive statistics:

- HIV-1 RNA (log<sub>10</sub> copies/mL)
- HIV-1 RNA categories (copies/mL): (a)  $\leq$  100,000, (b) > 100,000 to  $\leq$  400,000, and (c) > 400,000
- CD4+ cell count (/μL)
- CD4+ cell count categories (/ $\mu$ L): (a) < 50, (b)  $\geq$  50 to < 200, (c)  $\geq$  200 to < 350, (d)  $\geq$  350 to < 500, and (e)  $\geq$  500
- CD4 percentage (%)
- Mode of infection (HIV risk factors)
- HIV disease status
- eGFR<sub>CG</sub> (mL/min)
- Medical history: diabetes mellitus (Yes/No), hypertension (Yes/No), cardiovascular disease (Yes/No), and hyperlipidemia (Yes/No) (see Appendix 4 for details).
- HIV/HBV coinfection status (Yes/No/Missing, see Section 9.1 for definition)
- HIV/HCV coinfection status (Yes/No/Missing, see Section 9.2 for definition)

For categorical data, the CMH test (general association statistic for nominal data, and row means scores differ statistic for ordinal data) will be used to compare the 2 treatment groups. For continuous data, the 2-sided Wilcoxon rank sum test will be used to compare the 2 treatment groups.

# **5.3.** Medical History

General medical history data will be collected at screening and listed only. General medical history data will be coded using the current version of Medical Dictionary for Regulatory Activities (MedDRA).

### 6. EFFICACY ANALYSES

### 6.1. Primary Efficacy Endpoint

### 6.1.1. Definition of the Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm {U. S. Department of Health and Human Services 2015}. The proportions are expressed as percentages for presentation purposes.

# 6.1.2. US FDA-defined Snapshot Algorithm

The analysis window at Week 48 is defined as from Study Day 295 to Study Day 378, inclusive. All HIV-1 RNA data collected on-treatment (ie, data collected up to 1 day after permanent discontinuation of study drug or all available data for subjects who were still on study drug) will be used in the US FDA-defined snapshot algorithm. Virologic outcome will be defined as the following categories:

- **HIV-1 RNA < 50 copies/mL:** this includes subjects who have the last available on-treatment HIV-1 RNA < 50 copies/mL in the Week 48 analysis window
- HIV-1 RNA  $\geq$  50 copies/mL: this includes subjects
  - a) Who have the last available on-treatment HIV-1 RNA ≥ 50 copies/mL in the Week 48 analysis window, or
  - b) Who do not have on-treatment HIV-1 RNA data in the Week 48 analysis window and
    - 1) Who discontinue study drug prior to or in the Week 48 analysis window due to lack of efficacy, or
    - 2) Who discontinue study drug prior to or in the Week 48 analysis window due to reasons other than adverse event (AE), death, or lack of efficacy and have the last available on-treatment HIV-1 RNA ≥ 50 copies/mL
- No Virologic Data in the Week 48 Window: this includes subjects who do not have on-treatment HIV-1 RNA data in the Week 48 analysis window because of the following:
  - a) Discontinuation of study drug prior to or in the Week 48 analysis window due to AE or death (regardless of whether the last available on-treatment HIV-1 RNA < 50 copies/mL or not) or,
  - b) Discontinuation of study drug prior to or in the Week 48 analysis window due to reasons other than AE, death, or lack of efficacy and the last available on-treatment HIV-1 RNA < 50 copies/mL or,
  - c) Missing data during the window but on study drug.

The flowchart of the US FDA-defined snapshot algorithm is provided in Appendix 2.

The Week 48 virologic outcomes for the US FDA-defined snapshot algorithm will be listed.

## 6.1.3. Statistical Hypothesis for the Primary Efficacy Endpoint

**Null hypothesis:** The B/F/TAF group (Treatment Group 1) is at least 12% lower than the DTG + F/TAF group (Treatment Group 2) with respect to the proportion of subjects with HIV-1 RNA < 50 copies/mL ("response rate", as determined by the US FDA-defined snapshot algorithm) at Week 48.

**Alternative hypothesis:** The B/F/TAF group (Treatment Group 1) is less than 12% lower than the DTG + F/TAF group (Treatment Group 2) with respect to the proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48.

## 6.1.4. Primary Analysis of the Primary Efficacy Endpoint

The analysis purpose of the primary efficacy endpoint is to assess the noninferiority of treatment with B/F/TAF relative to treatment with DTG + F/TAF. Noninferiority will be assessed using a conventional 95% CI approach, with a noninferiority margin of 12%.

For each interim analyses performed for the IDMC at Weeks 12 and 24, an alpha of 0.00001 has been spent. Therefore, the significance level for the 2-sided test in the primary analysis at Week 48 will be 0.04998 (corresponding to 95.002% CI).

It will be concluded that B/F/TAF is noninferior to DTG + F/TAF if the lower bound of the 2-sided 95.002% CI of the difference (B/F/TAF group – DTG + F/TAF group) in the response rate is greater than -12%. The primary analysis will use the FAS.

The baseline stratum weighted difference in the response rate  $(P_1 - P_2)$  and its 95.002% CI will be calculated based on stratum-adjusted Mantel-Haenszel (MH) proportion as described as follows {Koch 1989}, where stratification factors include baseline HIV-1 RNA stratum ( $\leq 100,000 \text{ vs.} > 100,000 \text{ copies/mL}$ ) and region stratum (US vs. Ex-US):

$$P_1 - P_2 \pm Z_{(1-\alpha/2)} * SE(P_1 - P_2),$$

where

- $(P_1 P_2) = \frac{\sum w_h d_h}{\sum w_h}$ , is the stratum-adjusted MH proportion difference, where  $d_h = p_{1h} p_{2h}$  is the difference in the response rate between of the Treatment Groups 1 and 2 in stratum h (h = 1 to 4).
- $w_h = \frac{n_{1h}n_{2h}}{n_{1h} + n_{2h}}$ , is the weight based on the harmonic mean of sample size per treatment group for each stratum where  $n_{1h}$  and  $n_{2h}$  are the sample sizes of the Treatment Groups 1 and 2 in stratum h.

• SE(P<sub>1</sub> - P<sub>2</sub>) = 
$$\sqrt{\frac{\sum w_h^2 \left[ \frac{p_{1h}^* (1 - p_{1h}^*)}{n_{1h} - 1} + \frac{p_{2h}^* (1 - p_{2h}^*)}{n_{2h} - 1} \right]}{\left(\sum w_h^*\right)^2}}, \text{ where } p_{1h}^* = \frac{m_{1h} + 0.5}{n_{1h} + 1} \text{ and }$$

 $p_{2h}^* = \frac{m_{2h} + 0.5}{n_{2h} + 1}$ .  $m_{1h}$  and  $m_{2h}$  are the number of subjects with HIV-1 RNA < 50 copies/mL in the Treatment Groups 1 and 2 in stratum h.

- $\alpha = 0.04998$  for this study
- $Z_{(1-\alpha/2)} = Z_{0.97501} = 1.9601$  is the 97.501<sup>th</sup> percentile of the normal distribution

Note that if the computed lower confidence bound is less than -1, the lower bound is defined as -1. If the computed upper confidence bound is greater than 1, the upper bound is defined as 1.

The number and percentage of subjects with HIV-1 RNA < 50 copies/mL, HIV-1 RNA ≥ 50 copies/mL, and reasons for no virologic data at Week 48 will be summarized.

If noninferiority of B/F/TAF versus DTG + F/TAF is established, the same 95.002% CI used in evaluating noninferiority at Week 48 will be used to evaluate superiority. If the lower bound of the 95.002% CI is greater than 0, then superiority of B/F/TAF over DTG + F/TAF is established. The stratified 2-sided CMH test will also be used to assess superiority as a secondary assessment, where baseline stratum include baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US). The FAS will be used for the primary efficacy endpoint analysis and the superiority evaluation.

Additionally, the current study will be combined with study GS-US-380-1489, a Phase 3 study with a similar design to compare B/F/TAF with a FDC of abacavir (ABC) 600 mg / dolutegravir (DTG) 50 mg / lamivudine (3TC) 300 mg (ABC/DTG/3TC), to assess the superiority of B/F/TAF over ABC/DTG/3TC or DTG + F/TAF.

## 6.1.5. Secondary Analysis of the Primary Efficacy Endpoint

A secondary analysis based on the Week 48 PP analysis set will also be performed to evaluate the robustness of the primary analysis of the primary endpoint. The same adjusted alpha level 0.04998 (corresponding to 95.002% CI) will be used for this analysis.

In addition, the following analyses will be performed using the FAS to evaluate the interaction between region and treatment to assess homogeneity of treatment effect across different regions.

A region is defined as multiple sites combined based on geographical locations (see Appendix 3 for the region definition).

For each region, the difference in the proportion of subjects with HIV-1 RNA < 50 copies/mL between treatment groups and its 95% CI will be calculated based upon baseline HIV-1 RNA ( $\leq 100,000 \text{ vs.} > 100,000 \text{ copies/mL}$ ) stratum-adjusted MH proportion.

The CMH analysis will be used to estimate the odds ratio and corresponding 95% CI for each region and overall. The homogeneity of the odds ratios across different regions will be tested using a Breslow-Day test and a corresponding p-value will be reported.

As for adjusting randomization stratification for other stratified analyses, region stratum (US vs. Ex-US) will be used.

# 6.1.6. Subgroup Analysis of the Primary Efficacy Endpoint

The analysis of virologic response (HIV-1 RNA < 50 copies/mL, US FDA-defined snapshot algorithm) at Week 48 will be performed within each subgroup specified in Section 3.4 based on the FAS.

All subgroup analyses will be conducted using the US FDA-defined snapshot algorithm described in Section 6.1.2, adjusting for baseline HIV-1 RNA stratum ( $\leq 100,000 \text{ vs.} > 100,000 \text{ copies/mL}$ ) and region stratum (US vs. Ex-US), provided that they are not the factors defining the subgroup. For each level of subgroup factors, the proportion difference between the 2 treatment groups and 95% CIs will be computed based on the MH proportions adjusted by baseline HIV-1 RNA stratum ( $\leq 100,000 \text{ vs.} > 100,000 \text{ copies/mL}$ ) and region stratum (US vs. Ex-US), provide that they are not the factor defining the subgroup.

If the sample size in a subgroup is too small to calculate the proportion difference between 2 treatment groups and 95% CIs based on the stratum-adjusted MH proportions, then they will be computed based on normal approximation without stratification.

Additionally, a logistic regression model will be performed which includes the baseline stratification factor(s), subgroup factor, treatment, and treatment by subgroup factor. The baseline stratification factor(s) will include baseline HIV-1 RNA stratum ( $\leq 100,000 \text{ vs.} > 100,000 \text{ copies/mL}$ ) when analyzing region subgroup, region stratum (US vs. Ex-US) when analyzing baseline HIV-1 RNA subgroup, and both baseline HIV-1 RNA stratum ( $\leq 100,000 \text{ vs.} > 100,000 \text{ copies/mL}$ ) and region stratum (US vs. Ex-US) when analyzing other subgroups. The odds ratio and the associated 95% CI will be estimated within each subgroup. The homogeneity of the treatment effects between subgroups will be evaluated using a Wald test based on the interaction between treatment and the subgroup factor.

A forest plot of the treatment differences in HIV-1 RNA < 50 copies/mL (US FDA-defined snapshot algorithm) at Week 48 and their associated 95% CIs for each subgroup will be generated.

# 6.2. Secondary Efficacy Endpoints

## 6.2.1. Definition of the Secondary Efficacy Endpoints

The secondary efficacy endpoints include:

- The proportion of subjects with HIV-1 RNA < 50 copies/mL at Weeks 96 and 144 as determined by the US FDA-defined snapshot algorithm
- The proportion of subjects with HIV-1 RNA < 20 copies/mL at Weeks 48, 96 and 144 as determined by the US FDA-defined snapshot algorithm
- The change from baseline in log<sub>10</sub> HIV-1 RNA and CD4+ cell count at Weeks 48, 96, and 144

The secondary efficacy endpoints at future time points, such as Weeks 96 and 144, will not be summarized for the Week 48 interim analysis.

### 6.2.2. Analysis of the Secondary Efficacy Endpoints

6.2.2.1. Analysis of the Proportion of Subjects with HIV-1 RNA < 20 copies/mL as Determined by US FDA-defined Snapshot Algorithm

The proportion of subjects with HIV-1 RNA < 20 copies/mL at Week 48 will also be analyzed by the US FDA-defined snapshot algorithm based on FAS, except that CIs will be constructed at the 95% level.

6.2.2.2. Analysis of Log<sub>10</sub> HIV-1 RNA copies/mL and CD4+ Cell Count

All log<sub>10</sub> HIV-1 RNA data will be summarized using observed values (ie, missing will be excluded). While CD4+ cell count will be summarized using observed, on-treatment data (ie, data collected up to 1 day after permanent discontinuation of study drug or all available data for subjects who were still on study drug) for subjects in the FAS.

The changes from baseline in log10 HIV-1 RNA and CD4+ cell count at Week 48 will be summarized by treatment group using descriptive statistics. The differences in changes from baseline in log10 HIV-1 RNA and CD4+ cell count between the 2 treatment groups and the associated 95% CI will be constructed using analysis of variance (ANOVA) models, including treatment group, baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL), and region stratum (US vs. Ex-US) as fixed effects. The change from baseline in log10 HIV-1 RNA and CD4+ cell count will also be summarized at visits other than Week 48 by treatment group.

The change from baseline in CD4+ cell counts will also be analyzed based on the Week 48 PP analysis set.

The mean and 95% CI of change from baseline in log<sub>10</sub> HIV-1 RNA and CD4+ cell count over time will be plotted for the FAS.

In addition, the change from baseline in CD4+ cell counts with missing values imputed using the last observation carried forward (LOCF) method will be summarized at each visit based on the FAS. The algorithm for LOCF is as follows:

- If a value is missing in an analysis visit window, the missing value will be replaced with the
  last on-treatment value (ie, data collected up to 1 day after permanent discontinuation of
  study drug or all available data for subjects who were still on study drug) observed before the
  analysis visit window that has the missing value.
- Baseline values will be carried forward to impute the postbaseline value at a specific visit, if
  there is no nonmissing postbaseline observation collected prior to that visit.
- 6.3. Tertiary Efficacy Endpoints
- 6.3.1. Definition of the Tertiary Efficacy Endpoints



- 6.3.2. Analysis of the Tertiary Efficacy Endpoints
- 6.3.2.1. Analysis of the Proportion of Subjects with HIV-1 RNA < 50 copies/mL by Missing = Failure and Missing = Excluded Approaches







# 6.4. Changes From Protocol-Specified Efficacy Analyses

No change from the protocol-specified efficacy analysis is planned.

#### 7. SAFETY ANALYSES

Safety data will be summarized for the subjects in the safety analysis set. All safety data collected up to 30 days after permanent discontinuation of study drug and all available data for subjects who were still on study drug will be summarized by treatment group, unless specified otherwise. All safety data will be included in data listings.

#### 7.1. Adverse Events and Deaths

# 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using the current version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lowest-level term (LLT) will be provided in the AE dataset.

### 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) or Grade 4 (life threatening) according to toxicity criteria specified in the protocol. The severity grade of events for which the investigator did not record severity will be left as "missing" for data listings.

### 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE eCRF to the question of "Related to Study Treatment." Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if AEs met the definitions of SAE specified in the study protocol. Serious adverse events captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Drug Safety and Public Health (DSPH) Department before data finalization.

### 7.1.5. Treatment-Emergent Adverse Events

#### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of the study drug, or
- Any AEs leading to premature discontinuation of study drug.

## 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent if both of the following 2 criteria are met:

- The month and year (or year) of the AE onset is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The month and year (or year) of the AE onset is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date marked as ongoing or on or after the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

#### 7.1.6. Summaries of Adverse Events and Death

The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, HLT, PT, and treatment group. For other AEs described below, summaries will be provided by SOC, PT, and treatment group using the safety analysis set:

- Any Grade 2, 3, or 4 treatment-emergent AEs
- Any Grade 3 or 4 treatment-emergent AEs
- All treatment-emergent study drug-related AEs
- Any Grade 2, 3, or 4 treatment-emergent study drug-related AEs
- Any Grade 3 or 4 treatment-emergent study drug-related AEs
- All treatment-emergent SAEs
- All treatment-emergent study drug-related SAEs
- All treatment-emergent AEs that caused premature discontinuation from study drug

A brief, high-level summary of AEs described above will be provided by treatment group and by the number and percentage of subjects who experienced the above AEs. Treatment-emergent deaths observed in the study will be also included in this summary.
Treatment-emergent death refers to deaths that occurred between the first dose date and the last dose date plus 30 days (inclusive).

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC and HLT within each SOC (if applicable), and then by PT in descending order of total frequency within each SOC. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition to the above summary tables, all treatment-emergent AEs, Grade 3 or 4 treatment-emergent AEs, treatment-emergent study drug-related AEs, Grade 2, 3, or 4 treatment-emergent study drug-related AEs, and treatment-emergent SAEs will be summarized by PT only, in descending order of total frequency.

In addition, data listings will be provided for the following:

- All AEs
- Grade 3 and 4 AEs
- SAEs
- Study Drug-Related SAEs
- Deaths report
- AEs leading to premature discontinuation of study drug

#### 7.1.7. Additional Analysis of Adverse Events

#### 7.1.7.1. Stage 3 Opportunistic Illnesses in HIV

On an ongoing basis, AEs will be reviewed for events that might meet the definition of stage 3 opportunistic illnesses in HIV that are indicative of an AIDS-defining diagnoses (see Protocol Appendix 6). The Gilead medical monitor will review the possible stage 3 opportunistic illnesses and approve the events that meet the definition. Events that meet the stage 3 opportunistic illness definition of an AIDS-Defining Diagnosis will be listed.

#### 7.1.7.2. Cardiovascular or Cerebrovascular Events

Preferred terms for defining cardiovascular or cerebrovascular events are from relevant Standardised MedDRA Query (SMQ). The selected PT listing was provided by Gilead DSPH and reviewed by Gilead medical monitors, which is the same PT listing used to search "Cardiovascular Disease" medical history (see details in Appendix 4).

The number and percentage of subjects with treatment-emergent cardiovascular or cerebrovascular events and serious cardiovascular or cerebrovascular events by PT will be summarized by treatment group based on the safety analysis set. Statistical comparisons of the subject incidence rates between the 2 treatment groups will be performed using Fisher's exact test. A data listing of cardiovascular or cerebrovascular events will be provided.

### 7.1.7.3. Hepatic Events

Preferred terms for defining hepatic events are from 15 relevant SMQs, which are identified as non-infectious and non-congenital hepatobiliary disorders. The selected PT listing was provided by Gilead DSPH and reviewed by Gilead medical monitors (see details in Appendix 5).

The number and percentage of subjects with treatment-emergent hepatic events and serious hepatic events by PT will be summarized by treatment group based on the safety analysis set. Statistical comparisons of the subject incidence rates between the 2 treatment groups will be performed using Fisher's exact test. A data listing of hepatic events will be provided.

# 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the Safety Analysis Set. The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7.

A by-subject listing for laboratory test results will be provided by subject ID number and visit in chronological order for hematology, serum chemistry, and urinalysis separately. Values falling outside of the reference range and/or having a severity grade of 1 or higher on the Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities will be flagged in the data listings, as appropriate.

#### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by treatment group for each laboratory test specified in the study protocol as follows:

- Baseline values
- Values at each postbaseline analysis window
- Change from baseline at each postbaseline analysis window
- Percentage change from baseline to each postbaseline analysis window (if specified)

A baseline laboratory value will be defined as the last nonmissing value obtained on or prior to the date of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; SD values will be displayed to the reported number of digits plus 1.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

#### **Calcium Corrected for Albumin**

Calcium corrected for albumin will be calculated and summarized for the study. The following formula will be used when both serum calcium and albumin results for a given blood drawn are available and serum albumin value is < 4.0 g/dL.

• Calcium corrected for albumin (mg/dL) = serum calcium (mg/dL) +  $0.8 \times (4.0 - \text{albumin (g/dL)})$ 

Toxicity grading for calcium will be applied based on the corrected values.

#### **Estimated GFR**

The following formula will be used to calculate eGFR<sub>CG</sub>:

• eGFR<sub>CG</sub> (mL/min) =  $[(140 - age (yrs)) \times weight (kg) \times (0.85 \text{ if female})] / (SCr (mg/dL) \times 72)$ , where weight is total body mass in kilograms, and SCr is serum creatinine.

#### 7.2.2. Graded Laboratory Values

The Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities will be used for assigning toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately.

If there is any laboratory toxicity grading scale overlapping with the normal reference ranges (eg, grade 1 scale overlaps with normal reference ranges), laboratory values that are within the normal range will be grade 0, except for lipid tests.

For triglycerides, LDL, and cholesterol, the protocol-specified toxicity grading scale is for fasting test values, so nonfasting lipid results (or lipid results without a known fasting status) will not be graded or summarized by toxicity grades.

For the International normalized ratio (INR) of prothrombin time (PT), protocol-specified toxicity grade scale depends on the upper limit of normal range (ULN). While the ULN of INR depends on whether the subject is taking anticoagulant medication or not (ie, Not taking oral anticoagulant: 0.8 - 1.2; Taking oral anticoagulant: 2.0 - 3.0), this information is not collected by the reference laboratory. As a result, INR will be graded by assuming the subject is not taking

an oral anticoagulant, which is a conservative approach that may lead to over-reporting of abnormalities for INR. Consequently, INR and PT will not be included in summaries of laboratory abnormalities, but will be included in listings for the following reasons: 1) INR and PT are reflexive tests; 2) only the absolute values, not the toxicity grade, are needed for subject management purposes; and 3) more importantly, the toxicity grades for INR may be over-reported.

#### 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to 30 days after permanent discontinuation of study drug or the last available date for subjects who were still on study drug at the time of an interim analysis. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment-emergent.

Fasting glucose and nonfasting glucose (including glucose results without a known fasting status) are graded based on different grading scales as specified in the protocol. Treatment-emergent laboratory abnormalities will be summarized for fasting glucose. Maximum postbaseline grade, instead of treatment-emergent grade, for nonfasting glucose (including glucose results without a known fasting status) will be summarized, as nonfasting glucose was not assessed at baseline visit for most of the subjects; therefore, an abnormality is treatment-emergent or not cannot be determined for these subjects.

Both urine RBC based on microscopic examination, labeled as Hematuria (Quantitative), and urine blood based on a dipstick, labeled as Hematuria (Dipstick), are assessed routinely and assigned a toxicity grade in this study. Urine RBC based on microscopic examination will be presented in laboratory toxicity summary tables and listings while urine blood based on a dipstick will be presented in the listings only.

# 7.2.2.2. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Treatment-emergent laboratory abnormalities
- Treatment-emergent Grade 3 and 4 laboratory abnormalities
- Treatment-emergent Grade 2, 3 and 4 laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with any nonmissing postbaseline values up to 30 days after last dosing date.

A by-subject listing of all treatment-emergent laboratory abnormalities and treatment-emergent Grade 3 or 4 laboratory abnormalities will be provided by subject ID number and visit in chronological order.

## 7.2.3. Metabolic Laboratory Evaluations

For metabolic assessments, including fasting glucose and the lipid panel (ie, total cholesterol, triglycerides, LDL, HDL, total cholesterol to HDL ratio), only those measurements under fasting status will be summarized. P-values comparing the difference between the 2 treatment groups in baseline values and the change from baseline in metabolic assessment will be estimated from a 2-sided Wilcoxon rank sum test.

In addition, the number and percentage of subjects who took lipid modifying medications at study entry and initiated the medications during the study will be provided, respectively. Statistical comparisons of the subject incidence rates between the 2 treatment groups will be performed using Fisher's exact test.

A lipid modifying medication is defined as a medication with drug class = "LIPID MODIFYING AGENTS" and CMDECOD containing the wording of "STATIN".

A sensitivity analysis of fasting lipid tests will be performed by excluding subjects who took lipid modifying medications at study entry or initiated the medications during the study: baseline values, Week 48 values, and changes from baseline values at Week 48 will be summarized by treatment group using descriptive statistics. Baseline and change from baseline at Week 48 will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test. Only subjects with both baseline and Week 48 postbaseline values will be included in the analysis.

Median (Q1, Q3) of change from baseline in fasting metabolic assessments over time will be plotted by treatment group.

#### 7.2.4. Liver-Related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements:

- Aspartate aminotransferase (AST): (a)  $> 3 \times ULN$ , (b)  $> 5 \times ULN$ , (c)  $> 10 \times ULN$ , (d)  $> 20 \times ULN$
- Alanine aminotransferase (ALT): (a) > 3 × ULN, (b) > 5 × ULN, (c) > 10 × ULN,
   (d) > 20 × ULN
- AST or ALT: (a)  $> 3 \times ULN$ , (b)  $> 5 \times ULN$ , (c)  $> 10 \times ULN$ , (d)  $> 20 \times ULN$
- Total bilirubin: (a)  $> 1 \times ULN$ , (b)  $> 2 \times ULN$
- Alkaline phosphatase (ALP)  $> 1.5 \times ULN$
- AST or ALT >  $3 \times \text{ULN}$  and total bilirubin: (a) >  $1.5 \times \text{ULN}$ , (b) >  $2 \times \text{ULN}$
- AST or ALT > 3 × ULN and total bilirubin > 2 × ULN and ALP < 2 × ULN

The summary will include data from all postbaseline visits up to 30 days after the last dose of study drug. For individual laboratory tests, subjects will be counted once based on the most severe postbaseline value. For both the composite endpoint of AST or ALT and total bilirubin, and the composite endpoint of AST or ALT, total bilirubin, and ALP, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the safety analysis set with nonmissing postbaseline value of the tests in evaluation at the same postbaseline visit date.

Subjects with AST or ALT  $> 3 \times$  ULN will also be listed.

In addition, baseline, postbaseline, and change from baseline in AST, ALT, ALP, and total bilirubin will be summarized by treatment group and visit using descriptive statistics. Baseline and change from baseline will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test.

In addition, ALT flare, defined as subjects with ALT elevation > 2 x Baseline ALT and > 10 x ULN and confirmed at two consecutive visits, will be evaluated and listed for subjects with HIV/HBV coinfection at baseline.

#### 7.2.5. Renal-Related Laboratory Evaluations

#### 7.2.5.1. Serum Creatinine and eGFR<sub>CG</sub>

Baseline, postbaseline, and change from baseline in serum creatinine and  $eGFR_{CG}$  will be summarized by treatment group and visit using descriptive statistics. Baseline and change from baseline will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test.

Median (Q1, Q3) of change from baseline in serum creatinine and eGFR<sub>CG</sub> over time will be plotted by treatment group.

#### 7.3. Body Weight, Height, and Vital Signs

Descriptive statistics will be provided by treatment group for vital signs and body weight as follows:

- Baseline values
- Values at each postbaseline analysis window
- Change from baseline to each postbaseline analysis window

A baseline value will be defined as the last nonmissing value obtained on or prior to the date of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.

A by-subject listing of vital signs will be provided by subject ID number and visit in chronological order. In the same listing, a by-subject listing of body weight, height, and BMI will be provided.

#### 7.4. Prior and Concomitant Medications

# 7.4.1. Nonstudy Drug Antiretroviral Medications

Any nonstudy drug ARV medications used prior to, during, or after the study (if collected) will be coded using the Gilead-modified World Health Organization (WHO) Drug Dictionary for ARV medications. The WHO preferred name and drug code will be attached to the clinical database. All nonstudy drug ARV medications will be listed. No inferential statistics will be provided.

#### 7.4.2. Concomitant Non-ARV Medications

Concomitant non-ARV medications (ie, medications other than study drug that are taken while receiving study drug) will be coded using the WHO Drug Dictionary. The WHO preferred name and drug code will be attached to the clinical database. Use of concomitant medications from Study Day 1 up to the date of last dose of study drug will be summarized (number and percentage of subjects) by treatment group, WHO drug class and preferred name. Multiple drug use (by preferred name) will be counted only once per subject. The summary will be sorted alphabetically by drug class and then by decreasing total frequency within a class.

If the start or stop date of non-ARV medications is incomplete, the month and year (or year alone, if month is not recorded) of the start or stop date will be used to determine whether the non-ARVs are concomitant or not. The medication is concomitant if the month and year of the start or stop (or year of the start or stop, if month is not recorded) of the medication does not meet either of the following criteria:

- The month and year of start of the medication is after the date of the last dose of study drug
- The month and year of stop of the medication is before the date of the first dose of study drug

If the start and stop date of non-ARV medications are complete, the start date is not after last dose date and the stop date is not before first dose date, or the non-ARV medications are marked as ongoing and start date is on or before last dose date, the non-ARV medications are concomitant.

Summaries of non-ARV concomitant medications will be provided for the safety analysis set. Subjects with any non-ARV concomitant medications will be listed. No inferential statistics will be provided.

# 7.5. Electrocardiogram Results

A shift table of the investigators' assessment of ECG results at each scheduled postbaseline visit compared with baseline values will be presented by treatment group using the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant; or missing. The number and percentage of subjects in each cross-classification group of the shift table will be presented. Subjects with a missing value at baseline or postbaseline will not be included in the denominator for percentage calculation. No inferential statistics will be provided.

A by-subject listing for ECG assessment results will be provided by subject ID number and visits in chronological order.

#### 7.6. Other Safety Measures

A data listing will be provided for subjects experiencing pregnancy during the study. Physical examination data was not collected in the eCRF. Therefore, it will not be included in the analysis.

# 7.7. Changes From Protocol-Specified Safety Analyses

No change from the protocol-specified safety analysis is planned.

#### 8. PHARMACOKINETIC ANALYSES

Pharmacokinetic parameters will be computed for all subjects in the PK substudy analysis set. Only analytes from B/F/TAF group presented in Table 8-1 will be analyzed and evaluated.

Table 8-1. Treatment and Associated Analytes

| Treatment | Analyte |
|-----------|---------|
| | BIC |
| B/F/TAF | FTC |
| | TAF |

PK parameters to be estimated and analyzed in this substudy are listed and defined in PK abbreviations.

#### 8.1. Estimation of Pharmacokinetic Parameters

Pharmacokinetic parameters will be estimated by application of a nonlinear model using standard noncompartmental methods (WinNonlin® software). The linear up/log down trapezoidal rule will be used in conjunction with the appropriate noncompartmental model (usually input Model 200 for oral dosing), with input values for dose, time of dose, plasma concentration, and corresponding real time values, based on drug dosing times whenever possible.

All predose sample times of less than time zero will be converted to zero. Samples below the limit of quantitation of the bioanalytical assays that occur prior to the achievement of the first quantifiable concentration will be assigned a concentration value of zero to prevent overestimation of the initial AUC. Samples that are BLQ at all other time points will be treated as missing data. The nominal time point for a key event or dosing interval (tau) may be used to permit direct calculation of AUC over specific time intervals. The appropriateness of this approach will be assessed by the pharmacokineticist on a profile-by-profile basis.

Accurate estimation of several PK parameters, such as  $\lambda_z$  and  $t_{1/2}$ , are dependent on the accurate estimation of the terminal elimination phase of the drug. The appropriateness of calculating these parameters will be evaluated upon inspection of PK data on a profile-by-profile basis by the pharmacokineticist.

# 8.2. Analysis for Intensive PK (PK Substudy Analysis Set)

Plasma concentration will be listed for all subjects and summarized by nominal time point for subjects in the PK substudy analysis set.

PK parameters estimated for each analyte will be listed for all subjects and summarized for subjects in the PK substudy analysis set.

The descriptive statistics (n, mean, SD, coefficient of variation [%CV], minimum, median, maximum, Q1, Q3, geometric mean, and its 95% CI) will be presented for plasma concentration and parameter data. For concentration values BLQ, the number of subjects with values of BLQ will be presented. For PK parameter data, the mean and SD of the natural-log transformed values will be presented in addition to the summaries mentioned above.

The following tables, figures and listings (TFLs) will be provided for the intensive PK analysis for each analyte for subjects in the PK substudy analysis set:

- Table with individual subject concentration and summary statistics at each time point for each analyte
- Table with individual subject PK parameters and summary statistics for each analyte
- Mean (SD) concentration vs. time figures linear and semi-log plots for each analyte
- Median (Q1, Q3) concentration vs. time figures linear and semi-log plots for each analyte
- Individual plasma concentration vs. time figures linear and semi-log plots for each analyte
- Listing of the time points used in the calculation of the terminal elimination rate constant,  $\lambda_Z$ , for each analyte
- Listing of PK sampling details by subject including deviations in scheduled and actual draw times and procedures, individual blood sampling time deviations in minutes.
- Listing of study drug administration record for intensive PK dosing

#### 8.3. Analysis for Trough and Postdose PK (PK Analysis Set)

Only PK plasma samples collected through October 20<sup>th</sup>, 2016 were analyzed and their concentration data are available in the Week 48 interim analysis. The following listings will be provided for trough and postdose PK analysis for subjects in the PK analysis set:

- Listing of PK sampling details (PK samples collected as "Predose" during intensive PK collection or "Trough" PK samples [defined as samples collected within a range of 20.0 to 28.0 hours, inclusive, after previous dosing time] will be marked in the listing).
- Listing of study drug administration record for PK dosing.

PK sampling details for the intensive PK, trough PK, and postdose PK samples will be included in one listing. Similarly, study drug administration records for the intensive PK, trough PK, and postdose PK samples will also be included in one listing.

#### 8.4. Changes from Protocol-Specified Pharmacokinetic Analysis

No change from the protocol-specified PK analyses is planned.

#### 9. SPECIAL POPULATION ANALYSES

# 9.1. Analyses for HIV/HBV Coinfected Subjects

Subjects with HIV/HBV coinfection at baseline are defined as subjects meet any of the following two criteria:

- Positive HBsAg on or prior to the first dose date, or
- Negative HBsAg, negative HBsAb, positive HBcAb, and quantifiable HBV DNA (ie, HBV DNA ≥ 20 IU/mL) on or prior to the first dose date.

The following analyses will be conducted by treatment and overall for subjects with HIV/HBV coinfection at baseline:

- The proportion of subjects with HBV DNA < 29 IU/mL at baseline and Week 48 by missing = excluded approach.
- The change from baseline in log<sub>10</sub> HBV DNA (log<sub>10</sub> IU/mL)
- Treatment-emergent adverse events overall summary
- Treatment-emergent adverse events by SOC, HLT, and PT
- Treatment-emergent laboratory abnormalities
- The change from baseline for liver-related laboratory tests, including ALT, AST, ALP, GGT, total bilirubin, direct and indirect bilirubin.
- Listing of adverse events
- Listing of liver-related laboratory tests and HBV DNA results

HBV DNA will be analyzed using observed, on-treatment data (ie, data collected up to 1 day after permanent discontinuation of study drug or all available data for subjects who were still on study drug) for subject in the FAS with HIV/HBV coinfection at baseline.

Subjects with incident HIV/HBV coinfection while on study drug (if any) are defined as subjects who are not HIV/HBV coinfected at baseline and meet any of the following criteria:

- Positive HBsAg after the first dose date and on or prior to the date of permanent discontinuation of study drug, or
- Negative HBsAg, negative HBsAb, positive HBcAb, and quantifiable HBV DNA
   (ie, HBV DNA ≥ 20 IU/mL) after the first dose date and on or prior to the date of permanent discontinuation of study drug, or

• Experience any of the following adverse events (ie, selected MedDRA PTs from the SMQ of "Liver Infections") after the first dose date and on or prior to the date of permanent discontinuation of study drug: Acute hepatitis B, Chronic hepatitis B, Congenital hepatitis B infection, Hepatitis B, Hepatitis B core antibody positive, Hepatitis B DNA assay positive, Hepatitis B surface antigen positive, Hepatitis B virus test positive.

The following listings will be provided for subjects with incident HIV/HBV coinfection while on study drug (if any):

- Listing of adverse events
- Listing of liver-related laboratory tests and HBV DNA results

#### 9.2. Analyses for HIV/HCV Coinfected Subjects

Subjects with HIV/HCV coinfection at baseline are defined as subjects with positive HCVAb and quantifiable HCV RNA (ie, HCV RNA  $\geq$  15 IU/mL) on or prior to the first dose date. The following analyses will be provided for subjects with HIV/HCV coinfection at baseline:

- Treatment-emergent adverse events overall summary
- Treatment-emergent adverse events by SOC, HLT, and PT
- Treatment-emergent laboratory abnormalities
- Listing of adverse events
- Listing of liver-related laboratory tests and HCV RNA results

Subjects with incident HIV/HCV coinfection while on study drug are defined as subjects who are not HIV/HCV coinfected at baseline and meet any of the following criteria:

- Positive HCVAb after the first dose date and on or prior to the date of permanent discontinuation of study drug with baseline HCVAb Negative or missing, or
- Quantifiable HCV RNA (ie, HCV RNA ≥ 15 IU/mL) after the first dose date and on or prior to the date of permanent discontinuation of study drug, or
- Experience any of the following adverse events (ie, selected MedDRA PTs from the SMQ of "Liver Infections") after the first dose date and on or prior to the date of permanent discontinuation of study drug: Acute hepatitis C, Chronic hepatitis C, Hepatitis C, Hepatitis C antibody positive, Hepatitis C RNA positive, Hepatitis C virus test positive.

The following listings will be provided for subjects with incident HIV/HCV coinfection while on study drug:

- Listing of adverse events
- Listing of liver-related laboratory tests and HCV RNA results

# 10. REFERENCES

- Koch GG, Carr GJ, Amara IA, Stokes ME, Uryniak TJ. Categorical Data Analysis. Chapter 13 in Berry, D.A. (ed.). Statistical Methodology in the Pharmaceutical Sciences. New York: Marcel Dekker, Inc., 1989:pp. 414-21.
- U. S. Department of Health and Human Services, Food and Drug Administration (FDA), Center for Drug Evaluation and Research (CDER). Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment. Guidance for Industry. Revision 1. November 2015.

# 11. SOFTWARE

SAS® Version 9.4 (SAS Institute Inc., Cary, NC.) is to be used for all programming of tables, listings, and figures.

nQuery Advisor® Version 6.0 (Statistical Solutions, Cork, Ireland.) is to be used for sample size and power calculation.

Phoenix WinNonlin® Version 6.4 (Certara USA, Inc., Princeton, NJ, USA.) is to be used for all PK analyses.

# 12. SAP REVISION

| Revision Date<br>(dd month, yyyy) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

# 13. APPENDICES

Appendix 2. Flowchart of US FDA-defined Snapshot Algorithm (for Naïve Trial)

Appendix 3. Region Definition
Appendix 4. Selected Medical History

Appendix 5. Hepatic Events

Appendix 6. Programming Specification

Appendix 1. Study Procedures Table

Appendix Table 1. Study Procedures Table (Blinded Phase)

| | | | | | | | | | | | Enc | d of | Weel | €, q | | | Post-<br>Week 144 <sup>e,r</sup> | End of<br>Blinded | | Early |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedures | Screening <sup>a</sup> | Day 1 <sup>b</sup> | 4 | 8 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 108 | 120 | 132 | 144 | Every Treatmen | Treatment | 30-Day<br>Follow-up <sup>p</sup> | Study<br>Drugs<br>DC <sup>c</sup> |
| Informed Consent | X | | | | | | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>f</sup> | X <sup>f</sup> |
| Complete/Symptom- Directed Physical Exam | X | X | $X^{d}$ | $X^{d}$ | $X^{d}$ | X | $X^{d}$ | X | $X^{d}$ | $X^{d}$ | $X^{d}$ | X | $X^d$ | $X^d$ | $X^d$ | X | X <sup>d</sup> | X | $X^{d,f}$ | $\mathbf{X}^{\mathrm{f}}$ |
| 12-Lead ECG (performed supine) | X | X | | | | X | | X | | | | X | | | | X | X <sup>w</sup> | X | | X |
| Questionnaires | | X | X | | X | | | X | | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | | | | | | | |
| Vital signs (blood pressure, pulse, respiration rate, and temperature), including Weight | X | Х | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>f</sup> | X <sup>f</sup> |
| Urine Pregnancy Test <sup>g</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum Pregnancy Test | X | | | | | | | | | | | | | | | | | | | |
| Chemistry Profile <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>f</sup> | $X^{f}$ |
| Metabolic Assessments <sup>i</sup> | | X | | | X | X | | X | | X | | X | | X | | X | X | X | | |
| Estimated Glomerular Filtration Rate | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | $X^{f}$ | X |
| Hematology Profile <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>f</sup> | X <sup>f</sup> |
| Plasma HIV-1 RNA | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CD4+ Cell Count | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Plasma & Urine Storage Sample | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X |

| | | | | | | | | End of Week <sup>e, q</sup> | | | | | | | | | Post-<br>Week 144 <sup>e,r</sup> | End of<br>Blinded | Early<br>Study |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedures | Screening <sup>a</sup> | Day 1b | 4 | 8 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 108 | 120 | 132 | 144 | Every<br>12 Weeks | Treatment<br>Visit | Drugs |
| HCV Serology <sup>u</sup> | X | | | | | | | X | | | | X | | | | X | X | | |
| HIV-1 Genotype <sup>k</sup> | X | | | | | | | | | | | | | | | | | | |
| HIV-1 Genotype/Phenotype <sup>e</sup> | 6 | | | | | | | | | | 2 3 | 8 | | | | Q 4 | | | Xe |
| Single PK Sample <sup>1</sup> | | | | X | | X | X | | | | | | | | | | | | |
| Trough and Post Dose PK Sample <sup>m</sup> | | | X | | X | | DC | | | | | | | | | | | | |
| Optional PPD | | X | | | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | | |
| Provide subject dosing diary to subjects | 5 7. | X | X | X | X | X | .d 6. | | | | 9 - 75 | 9 9 | | | | 9 75 | Lit C | | |
| Optional PK Substudy <sup>n</sup> | | | X | X | | | | | | | | | | | | | | | |
| Optional PBMC Substudy <sup>o</sup> | | X | | | | | X | | | | X | | | | X | | ru. | | |
| HBV blood panel | X | | | | $\mathbf{X}^{t}$ | $\mathbf{X}^{t}$ | r 6 | $X^{t}$ | | $\mathbf{X}^{t}$ | | $\mathbf{X}^{t}$ | | $\mathbf{X}^{t}$ | | $\mathbf{X}^{t}$ | X | | Š. |
| Plasma HBV DNA <sup>t</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Study Drug Dispensation | | $X^{b}$ | X | X | X | X | X | X | X | X | X | X | X | Х | X | X | X | Xs | |
| Study Drug Accountability | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

- a Evaluations to be completed within 30 days prior to Day 1.
- b Initiation of the first dose of study drug is to take place in-clinic following completion of study procedures at the Day 1 visit.
- c Early Study Drugs Discontinuation visit to occur within 72 hours of last dose of study drug. Subjects will be asked to continue attending the scheduled study visits through the End of Blinded Treatment Visit even if the subject discontinues study drug.
- d Symptom-directed physical examination as needed.
- e HIV-1 genotype and phenotype testing for subjects with virologic failure. Following virologic rebound, subjects will be asked to return to the clinic (2-3 weeks later) prior to the next scheduled visit or at the next scheduled study visit, for a HIV-1 RNA and HIV-1 genotype and phenotype (reverse transcriptase, protease and integrase genotype and phenotype) blood draw. Based on the results of this testing, subjects should be managed according to the Virologic Rebound Schema (Protocol Section 6.12).
- f Any adverse event or test showing abnormal results that is believed to have a possible or probable causal relationship with the study drug will be repeated weekly (or as often as deemed prudent by the Investigator) until the abnormality is resolved, returns to baseline, or is otherwise explained.
- g Females of childbearing potential only. Positive urine pregnancy tests will be confirmed with a serum test.

- h Chemistry profile: alkaline phosphatase, AST, ALT, GGT, total bilirubin, direct and indirect bilirubin, total protein, albumin, LDH, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid and amylase (reflex lipase testing is performed in subjects with total amylase > 1.5 x ULN). At Day 1, Weeks 12, 24, 48, 72, 96, 120 and 144, every 24 weeks post Week 144, and End of Blinded Treatment Visit, analyses of glucose will be done as part of the fasting metabolic assessments every 24 weeks and not as part of the chemistry profile. Additionally: TSH will be analyzed at Screening, Day 1, Weeks 24, 48, 72, 96,
- 120, and 144 followed by every 24 weeks post Week 144, End of Blinded Treatment Visit and Early Study Drugs Discontinuation visit. PT/INR to be performed at Day 1.

  i Fasting (no food or drinks, except water, at least 8 hours prior to blood collection) glucose and lipid panel (total cholesterol, HDL, direct LDL, triglycerides). If the subject has not fasted prior to the visit, the visit may proceed, but the subject must return within 72 hours in a fasted state to draw blood for the metabolic assessments.
- i CBC with differential and platelet count.
- k The Investigator must have received the results from the screening genotype report before proceeding with the Day 1 visit. Screening genotype report must show sensitivity to TFV and FTC. If genotype results from a local laboratory obtained ≤ 90 days prior to screening visit date show sensitivity to these drugs, this genotype will be acceptable to fulfill this inclusion criterion in the event that the genotype obtained at screening is not yet available and all other inclusion/exclusion criteria have been confirmed.
- 1 A single PK blood sample will be collected at any time pre or post-dose
- m A trough PK blood sample will be collected between 20-28 hours following the last dose. Following an observed dose, a single post dose blood sample will be collected between 1 and 4 hours post dose.
- n A pharmacokinetic (PK) substudy will be performed in a subset of subjects (n=30) at selected study sites. The PK substudy visit must occur at the Week 4 or Week 8 visits. The substudy will include intensive PK profiling in plasma.
- o A PBMC substudy will be performed in a subset of subjects (n=50) at selected study sites. A blood sample will be collected at Day 1, Weeks 36 84, and 132.
- p Only required for those subjects not enrolling in the open-label rollover extension, those subjects who prematurely discontinue study drugs and do not continue in the study through at least one subsequent visit after the Early Study Drugs Discontinuation Visit. For the purpose of scheduling a 30-Day Follow-Up Visit, a ± 6 days window may be used.
- q Study visits are to be completed within ± 2 days of the protocol-specified visit date based on the Day 1 visit through Week 12 and completed within ± 6 days through to Week 144, unless otherwise specified. The visit window at Weeks 48, 96, and 144 will be ± 6 weeks of the protocol-specified visit date.
- r After Week 144, all subjects will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Visit window of ± 6 days for study visits post Week 144.
- s Open label study drug, B/F/TAF FDC will be dispensed to subjects participating in the Open-Label Rollover extension for up to 48 weeks.
- t HBV blood panel will be performed at Screening (Hepatitis B virus surface antigen (HBsAg), Hepatitis B virus surface antibody (HBsAb) and Hepatitis B virus core antibody (HBcAb)). For subjects who meet the definition of HBV infection at any visit: The following will be conducted by the central laboratory: HBsAb, HBsAg (qualitative and quantitative) and HBeAg (if negative, reflex HBeAb) (Weeks 12, 24, 48, 72, 96 and every 24 weeks post Week 96) and Plasma HBV DNA (every visit). For subjects who do NOT meet the definition of HBV infection at any visit: The following will be conducted by the central laboratory: Hepatitis B surface antibody (HBsAb), Hepatitis B virus core antibody (HBsAb), and Hepatitis B virus surface antigen serology (HBsAg). Subjects who are HBsAg and/or HBcAb positive will have a reflex test for HBV DNA (viral load) (Week 48, 96 and 144 and every 48 weeks post Week 144)
- Hepatitis C virus (HCVAb) serology. Subjects who are HCVAb positive will have a HCV RNA test performed (Week 48, 96 and 144 and every 48 weeks post Week 144)
- v Randomization may be performed up to 3 days prior to the in-clinic Day 1 visit provided that all screening procedures have been completed and subject eligibility has been confirmed.
- w To be performed every 48 weeks.

# **Appendix Table 2.** Study Procedures Table (Open Label Rollover Extension)

| | End of Blinded | | End of | Week <sup>e,l</sup> | | 30-Day | Early Study Drugs |
|---|---|---|---|---|---|---|---|
| <b>Study Procedures</b> | Treatment Visit <sup>a</sup> | 12 OL | 24 OL | 36 OL | 48 OL | Follow-up <sup>k</sup> | DC <sup>c</sup> |
| Adverse Events | X | X | X | X | X | $X^{f}$ | $X^{f}$ |
| Concomitant Medications | X | X | X | X | X | X | X |
| Complete/Symptom-Directed Physical Exam | X | $X^{d}$ | X <sup>d</sup> | $X^d$ | X <sup>d</sup> | $X^{d,f}$ | <b>X</b> <sup>f</sup> |
| 12-Lead ECG (performed supine) | X | | | | | | |
| Vital signs (blood pressure, pulse, respiration rate, and temperature), including Weight | X | X | X | X | X | X | X |
| Urinalysis | X | X | X | X | X | $X^{\mathrm{f}}$ | $X^{f}$ |
| Urine Pregnancy Test <sup>g</sup> | X | X | X | X | X | X | X |
| Chemistry Profile <sup>h</sup> | X | X | X | X | X | $X^{\mathrm{f}}$ | X <sup>f</sup> |
| Metabolic Assessments <sup>i</sup> | X | | X | | X | | |
| Estimated Glomerular Filtration Rate | X | X | X | X | X | $X^{\mathrm{f}}$ | X |
| Hematology Profile <sup>i</sup> | X | X | X | X | X | $X^{\mathrm{f}}$ | X <sup>f</sup> |
| Plasma HIV-1 RNA | X | X | X | X | X | X | X |
| CD4+ Cell Count | X | X | X | X | X | X | X |
| Plasma & Urine Storage Sample | X | X | X | X | X | | X |
| HBV Blood Panel <sup>m</sup> | | | X <sup>m</sup> | | X <sup>m</sup> | | |
| Plasma HBV DNA <sup>m</sup> | | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> | | |
| HCV Serology <sup>n</sup> | | | | | X <sup>n</sup> | | |
| HIV-1 Genotype/Phenotype <sup>e</sup> | | | | | | | X <sup>e</sup> |

| | End of Blinded | | End of | Week <sup>e,l</sup> | | 30-Day | Early Study Drugs |
|---|---|---|---|---|---|---|---|
| <b>Study Procedures</b> | Treatment Visit <sup>a</sup> | 12 OL | 24 OL | 36 OL | 48 OL | Follow-up <sup>k</sup> | DC <sup>c</sup> |
| Study Drug Dispensation <sup>b</sup> | X <sup>b</sup> | X | X | X | | | |
| Study Drug Accountability | X | X | X | X | X | | X |

- a Once the last subject completes the Week 144 visit and Gilead completes the Week 144 analysis, all subjects will return to the clinic (within 30 days ± 6 days) for an End of Blinded Treatment Visit. At the End of Blinded Treatment Visit, if safety and efficacy of B/F/TAF FDC is demonstrated following review of unblinded data, subjects in a country where GS-9883/F/TAF FDC is not available, will be given the option to receive B/F/TAF FDC in an open label extension phase for up to 48 weeks, or until the product becomes accessible to subjects through an access program, or until Gilead Sciences elects to discontinue the study in that country, whichever occurs first.
- b Open label study drug, B/F/TAF FDC will be dispensed to subjects participating in the Open-Label Rollover extension for up to 48 weeks.
- c Subjects who discontinue study drug during the open label rollover extension portion of the study will be asked to return to the clinic within 72 hours of stopping study drugs for the Early Study Drugs Discontinuation Visit followed by a 30-Day Follow-Up Visit. The subject will not continue attending the scheduled study visits.
- d Symptom-directed physical examination as needed.
- e HIV-1 genotype and phenotype testing for subjects with virologic failure. Following virologic rebound, subjects will be asked to return to the clinic (2-3 weeks later) prior to the next scheduled visit or at the next scheduled study visit, for a HIV-1 RNA and HIV-1 genotype and phenotype (reverse transcriptase, protease, and integrase genotype and phenotype) blood draw. Based on the results of this testing, subjects should be managed according to the Virologic Rebound Schema (Protocol Section 6.12.1).
- f Any adverse event or test showing abnormal results that is believed to have a possible or probable causal relationship with the study drug will be repeated weekly (or as often as deemed prudent by the Investigator) until the abnormality is resolved, returns to Day 1, or is otherwise explained.
- g Females of childbearing potential only. Positive urine pregnancy tests will be confirmed with a serum test.
- h Chemistry profile: alkaline phosphatase, AST, ALT, GGT, total bilirubin, direct and indirect bilirubin, total protein, albumin, LDH, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid and amylase (reflex lipase testing is performed in subjects with total amylase > 1.5 x ULN). At Week 24 OL and Week 48 OL, and End of Blinded Treatment Visit, analyses of glucose will be done as part of the fasting metabolic assessments and not as part of the chemistry profile. For all subjects, TSH will be done at the End of Blinded Treatment Visit, Week 24 OL, Week 48 OL, and Early Study Drug Discontinuation Visit.
- Fasting (no food or drinks, except water, at least 8 hours prior to blood collection) glucose and lipid panel (total cholesterol, HDL, direct LDL, triglycerides) every 24 weeks. If the subject has not fasted prior to the visit, the visit may proceed, but the subject must return within 72 hours in a fasted state to draw blood for the metabolic assessments.
- i CBC with differential and platelet count.
- k Subjects who complete the open-label rollover extension will be required to return to the clinic 30 days after the completion of study drugs for the 30-Day Follow-Up Visit. Subjects who permanently discontinue study drugs during the open-label rollover extension will be asked to return to the clinic 30 days after the completion of the Early Study Drugs Discontinuation Visit for the 30-Day Follow-Up Visit. For the purpose of scheduling a 30-Day Follow-Up Visit, a ± 6 days window may be used.
- 1 Study visits are to be completed within ± 2 days of the protocol-specified visit date based on the End of Blinded Treatment Visit date through Week 12 OL and completed within ± 6 days of the protocol-specified visit date every 12 weeks thereafter, unless otherwise specified
- m For subjects who meet the definition of HBV infection at any visit: The following will be conducted by the central laboratory: HBsAb, HBsAg (qualitative and quantitative) and HBeAg (if negative, reflex HBeAb) (every 24 weeks) and Plasma HBV DNA (every 12 weeks). For subjects who do NOT meet the definition of HBV infection at any visit: The following will be conducted by the central laboratory: Hepatitis B surface antibody (HBsAb), Hepatitis B virus core antibody (HBcAb), and Hepatitis B virus surface antigen serology (HBsAg). Subjects who are HBsAg and/or HBcAb positive will have a reflex test for HBV DNA (viral load) (every 48 weeks throughout study including OL)
- n Hepatitis C virus (HCVAb) serology. Subjects who are HCVAb positive will have a HCV RNA test performed. (every 48 weeks)

# Appendix 2. Flowchart of US FDA-defined Snapshot Algorithm (for Naïve Trial)

The following flowchart for US FDA-defined snapshot algorithm is based on the US FDA Guidance on Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment {U. S. Department of Health and Human Services 2015}



<sup>\*</sup> On-treatment data include all data collected up to 1 day after permanent discontinuation of study drug or all available data for subjects who were still on study drug.

**Appendix 3.** Region Definition

| Region | Country Name | State | No. of Subjects in Safety<br>Analysis Set or FAS<br>(N=645) | Total No. of Subjects<br>by Region in Safety<br>Analysis Set or FAS<br>(N=645) |
|---|---|---|---|---|
| Danian 1 | AUSTRALIA (AUS) | | 14 | 35 |
| Region 1 | CANADA (CAN) | | 21 | |
| | BELGIUM (BEL) | | 8 | 179 |
| | FRANCE (FRA) | | 12 | |
| D 2 | GERMANY (DEU) | | 48 | |
| Region 2 | ITALY (ITA) | | 33 | |
| | SPAIN (ESP) | | 34 | |
| | UNITED KINGDOM (GBR) | | 44 | |
| D 2 | UNITED STATES (USA) | CA | 28 | 35 |
| Region 3 | UNITED STATES (USA) | WA | 7 | |
| | UNITED STATES (USA) | AZ | 9 | 90 |
| Region 4 | UNITED STATES (USA) | CO | 2 | |
| | UNITED STATES (USA) | TX | 79 | |
| | UNITED STATES (USA) | IL | 7 | 33 |
| | UNITED STATES (USA) | IN | 1 | |
| Region 5 | UNITED STATES (USA) | MI | 13 | |
| | UNITED STATES (USA) | MO | 11 | |
| | UNITED STATES (USA) | ОН | 1 | |
| | UNITED STATES (USA) | DC | 13 | 54 |
| | UNITED STATES (USA) | MA | 8 | |
| | UNITED STATES (USA) | MD | 1 | |
| Region 6 | UNITED STATES (USA) | NJ | 11 | |
| | UNITED STATES (USA) | NY | 10 | |
| | UNITED STATES (USA) | PA | 7 | |
| | UNITED STATES (USA) | VA | 4 | |
| | UNITED STATES (USA) | GA | 36 | 62 |
| Region 7 | UNITED STATES (USA) | NC | 25 | |
| | UNITED STATES (USA) | SC | 1 | |
| | DOMINICAN REPUBLIC (DOM) | | 45 | 157 |
| Region 8 | UNITED STATES (USA) | FL | 99 | |
| | UNITED STATES (USA) | PR* | 13 | |

<sup>\*</sup> PR = Puerto Rico.

Note: In general, a region is defined as multiple sites combined based on geographical locations. For example, for international studies, sites from each country or multiple neighboring counties were combined; and for US studies, sites from each state or multiple neighboring states were combined.

## **Appendix 4.** Selected Medical History

Number and percentage of subjects with selected medical history of Diabetes Mellitus, Hypertension, Cardiovascular Disease, and Hyperlipidemia will be summarized by treatment as baseline disease characteristics. A subject who had medical history of one of these diseases is a subject who experience at least one of the following events:

- At least 1 medical history record with MedDRA PT (mh.MDRPT) in the selected PT listing for the corresponding disease with start date on or prior to the first dose date.
- At least 1 adverse event record with MedDRA PT (ae.MDRPT) in the selected PT listing for the corresponding disease with start date on or prior to the first dose date.
- At least 1 concomitant medications record with medication class and indication in the following selected listing for the corresponding disease with start date on or prior to the first dose date.

If the start date is incomplete but the month and year (or year alone) of the start date is the same as or before the month and year (or year alone) of the first dosing date of study drug, then the event will be included. If the start date is completed missing, the event will be included.

Four variables (ie, DIABETES, HTENSION, CARDDIS, and HLIPDEM) will be added to raw Medical History and Adverse Events datasets. A medical history or an adverse event record will be flagged for a disease of interest if its MedDRA PT included in the pre-specified PT list for the corresponding disease of interest, which include all PTs from the narrow or broad search of the following SMQs under MedDRA 19.1 provided by Gilead DSPH and reviewed by Gilead medical monitors.

| Disease of Interest | SMQ Source |
|---|---|
| Diabetes Mellitus (DIABETES) | Hyperglycaemia/new onset diabetes mellitus (SMQ) – Narrow Scope Term |
| Hyperlipidemia (HLIPDEM) | Dyslipidaemia (SMQ) |
| Hypertension (HTENSION) | Hypertension (SMQ) |
| | Ischaemic central nervous system vascular conditions (SMQ) – Narrow Scope Term |
| Cardiovascular disease (CARDDIS) | Myocardial infarction (SMQ) - Narrow Scope Term |
| ( | Other ischaemic heart disease (SMQ) - Narrow Scope Term |

Similarly, four variables (ie, DIABETES, HTENSION, CARDDIS, and HLIPDEM) will be added to raw Concomitant Medication dataset. A concomitant medication record will be flagged for a disease of interest if its medication class and indication included in the following listing for the corresponding disease of interest.

The selected combination of medication class and indication are listed as follows, which was reviewed by Gilead medical monitors.

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| Нуре | rtension (HTENSION) | | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | | LISINOPRIL |
| 2 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ANTI-HYPERTENSIVE | LOSARTAN |
| 3 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPENTENSION | RAMIPRIL |
| 4 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | CAPTOPRIL |
| 5 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | ENALAPRIL |
| 6 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | HYDROCHLOROTHIAZIDE<br>W/OLMESARTAN |
| 7 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | OLMESARTAN MEDOXOMIL |
| 8 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | RAMIPRIL |
| 9 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | SALUTEC |
| 10 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | VALSARTAN |
| 11 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION<br>STAGE I | CAPTOPRIL |
| 12 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION<br>STAGE 1 | CANDESARTAN |
| 13 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | BENIGN ESSENTIAL<br>HYPERTENSION | LISINOPRIL |
| 14 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | BENIGN ESSENTIAL<br>HYPERTENSION | LOSARTAN |
| 15 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL<br>(PRIMARY)HYPERTESION | ZESTORETIC |
| 16 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | COROVAL B |
| 17 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | ENALAPRIL MALEATE |
| 18 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | LISINOPRIL |
| 19 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | LOSARTAN |
| 20 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | TRIBENZOR |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 21 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | ZESTORETIC |
| 22 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL PRIMARY<br>HYPERTENSION | IRBESARTAN |
| 23 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | COVERAM |
| 24 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | ENALAPRIL |
| 25 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | IRBESARTAN |
| 26 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | LISINOPRIL |
| 27 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | LOSARTAN |
| 28 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | LOSARTAN POTASSIUM |
| 29 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | RAMIPRIL |
| 30 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BOLD PRESSURE | LOSARTAN |
| 31 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HISTORY OF MYOCARDITIS | RAMIPRIL |
| 32 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HTN | ZESTORETIC |
| 33 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERRTENSION | ZESTORETIC |
| 34 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTEENSION | LISINOPRIL |
| 35 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | AMLODIPINE<br>W/HYDROCHLOROTHIAZIDE/V<br>ALSARTAN |
| 36 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | AMLODIPINE W/VALSARTAN |
| 37 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BENAZEPRIL |
| 38 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BENAZEPRIL<br>HYDROCHLORIDE |
| 39 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BENICAR HCT |
| 40 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BI PREDONIUM |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 41 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CANDESARTAN |
| 42 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CANDESARTAN CILEXETIL |
| 43 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CAPTOPRIL |
| 44 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CO-DIOVAN |
| 45 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | COROVAL B |
| 46 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | DIOVAN AMLO |
| 47 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | DIOVAN TRIPLE |
| 48 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | EDARBYCLOR |
| 49 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | ENALAPRIL |
| 50 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | ENALAPRIL MALEATE |
| 51 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | FOSINOPRIL |
| 52 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | HYDROCHLOROTHIAZIDE<br>W/LOSARTAN |
| 53 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | HYZAAR |
| 54 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | IRBESARTAN |
| 55 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | KARVEA HCT |
| 56 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | LISINOPRIL |
| 57 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | LOSARTAN |
| 58 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | LOSARTAN POTASSIUM |
| 59 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | NAPRIX A |
| 60 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | OLMESARTAN MEDOXOMIL |
| 61 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | PERINDOPRIL ERBUMINE |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 62 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | PRITORPLUS |
| 63 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | QUINAPRIL |
| 64 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | RAMIPRIL |
| 65 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | SALUTEC |
| 66 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | TELMISARTAN |
| 67 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | TRIBENZOR |
| 68 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | VALSARTAN |
| 69 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | VASERETIC |
| 70 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | ZESTORETIC |
| 71 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION ESSENTIAL | CANDESARTAN CILEXETIL |
| 72 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION ESSENTIAL | DIOVAN TRIPLE |
| 73 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, BENIGN | LISINOPRIL |
| 74 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, BILATERAL<br>LOWER LEG SWELLING | LISINOPRIL |
| 75 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, ESSENTIAL | ZESTORETIC |
| 76 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, WORSENING<br>HYPERTENSION | LISINOPRIL |
| 77 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSIONPROPHYLAXIS | RAMIPRIL |
| 78 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSIVE | RAMIPRIL |
| 79 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSIVE CRISIS | CAPTOPRIL |
| 80 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENTION | LISINOPRIL |
| 81 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTONIA | RAMIPRIL |
| 82 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPOKALEMIA | LOSARTAN POTASSIUM |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 83 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | POOR CONTROL OF BLOOD<br>PRESSURE | LISINOPRIL |
| 84 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PREVENTATIVE FOLLOWING<br>ACUTE MYCARDIAL<br>INFARCTION | PERINDOPRIL |
| 85 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PRIMARY ESSENTIAL<br>HYPERTENSION | ENALAPRIL MALEATE |
| 86 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PROTEINURIA | BENAZEPRIL |
| 87 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PROTEINURIA | ENALAPRIL |
| 88 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PROTEINURIA | LISINOPRIL |
| 89 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING HYPERTENSION | BENAZEPRIL |
| 90 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING HYPERTENSION | PERINDOPRIL |
| 91 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING HYPERTENSION | PRETERAX ARGININE |
| 92 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING OF<br>HYPERTENSION | LISINOPRIL |
| 93 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING OF<br>HYPERTENSION | RAMIPRIL |
| 94 | ANTIHYPERTENSIVES | BENIGN HIGH BLOOD<br>PRESSURE | DOXAZOSIN |
| 95 | ANTIHYPERTENSIVES | EXACERBATION OF<br>HYPERTENSION | CLONIDINE |
| 96 | ANTIHYPERTENSIVES | HEADACHE | HYDRALAZINE |
| 97 | ANTIHYPERTENSIVES | HIGH BLOOD PRESSURE | CLONIDINE HYDROCHLORIDE |
| 98 | ANTIHYPERTENSIVES | HIGH BLOOD PRESSURE | RILMENIDINE |
| 99 | ANTIHYPERTENSIVES | HYPERTENSION | CLONIDINE |
| 100 | ANTIHYPERTENSIVES | HYPERTENSION | CLONIDINE HYDROCHLORIDE |
| 101 | ANTIHYPERTENSIVES | HYPERTENSION | DOXAZOSIN |
| 102 | ANTIHYPERTENSIVES | HYPERTENSION | DOXAZOSIN MESILATE |
| 103 | ANTIHYPERTENSIVES | HYPERTENSION | HYDRALAZINE |
| 104 | ANTIHYPERTENSIVES | HYPERTENSION | HYDRALAZINE<br>HYDROCHLORIDE |
| 105 | ANTIHYPERTENSIVES | HYPERTENSION | METHYLDOPA |
| 106 | ANTIHYPERTENSIVES | HYPERTENSION | TADALAFIL |
| 107 | ANTIHYPERTENSIVES | PULMONARY HYPERTENSION | TADALAFIL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 108 | ANTIHYPERTENSIVES | VASODILATION-STENT<br>PROCEDURE | HYDRALAZINE |
| 109 | ANTIHYPERTENSIVES | WORSENING HYPERTENSION | HYDRALAZINE<br>HYDROCHLORIDE |
| 110 | BETA BLOCKING AGENTS | ARTERIAL HYPERTENSION | ATENOLOL |
| 111 | BETA BLOCKING AGENTS | ARTERIAL HYPERTENSION | METOPROLOL SUCCINATE |
| 112 | BETA BLOCKING AGENTS | ARTERIAL HYPERTENSION /<br>ICHEMIC HEART DISEASE | BISOPROLOL |
| 113 | BETA BLOCKING AGENTS | ESSENTIAL HYPERTENSION | METOPROLOL |
| 114 | BETA BLOCKING AGENTS | HEART FAILURE AND<br>HYPERTENSION | CARVEDILOL |
| 115 | BETA BLOCKING AGENTS | HEART HEALTH | ATENOLOL |
| 116 | BETA BLOCKING AGENTS | HIGH BLOOD PRESSURE | ATENOLOL |
| 117 | BETA BLOCKING AGENTS | HIGH BLOOD PRESSURE | BISOPROLOL<br>W/HYDROCHLOROTHIAZIDE |
| 118 | BETA BLOCKING AGENTS | HIGH BLOOD PRESSURE | METOPROLOL |
| 119 | BETA BLOCKING AGENTS | HISTORY OF MYOCARDITIS | BISOPROLOL |
| 120 | BETA BLOCKING AGENTS | HYPERTENSION | ATENOLOL |
| 121 | BETA BLOCKING AGENTS | HYPERTENSION | BISOPROLOL FUMARATE |
| 122 | BETA BLOCKING AGENTS | HYPERTENSION | CARVEDILOL |
| 123 | BETA BLOCKING AGENTS | HYPERTENSION | LABETALOL |
| 124 | BETA BLOCKING AGENTS | HYPERTENSION | METOPROLOL |
| 125 | BETA BLOCKING AGENTS | HYPERTENSION | METOPROLOL SUCCINATE |
| 126 | BETA BLOCKING AGENTS | HYPERTENSION | METOPROLOL TARTRATE |
| 127 | BETA BLOCKING AGENTS | HYPERTENSION | NEBICARD V |
| 128 | BETA BLOCKING AGENTS | HYPERTENSION | NEBICARD-H |
| 129 | BETA BLOCKING AGENTS | HYPERTENSION | NEBIVOLOL |
| 130 | BETA BLOCKING AGENTS | HYPERTENSION | NEBIVOLOL HYDROCHLORIDE |
| 131 | BETA BLOCKING AGENTS | HYPERTENSION | PROPRANOLOL |
| 132 | BETA BLOCKING AGENTS | HYPERTENSION | PROPRANOLOL<br>HYDROCHLORIDE |
| 133 | BETA BLOCKING AGENTS | HYPERTENSION AND MIGRAINE | ATENOLOL |
| 134 | BETA BLOCKING AGENTS | HYPERTENSION ESSENTIAL | ATENOLOL |
| 135 | BETA BLOCKING AGENTS | HYPERTENTION | METOPROLOL SUCCINATE |
| 136 | BETA BLOCKING AGENTS | HYPETENSION | BISOPROLOL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 137 | BETA BLOCKING AGENTS | PAROXYSM OF SINUS<br>TACHYCARDIA | PROPRANOLOL |
| 138 | BETA BLOCKING AGENTS | PRIMARY ESSENTIAL<br>HYPERTENSION | CARVEDILOL |
| 139 | BETA BLOCKING AGENTS | RAPID HEART BEAT | METOPROLOL SUCCINATE |
| 140 | CALCIUM CHANNEL BLOCKERS | ANTIHYPERTENSIVE | AMLODIPINE |
| 141 | CALCIUM CHANNEL BLOCKERS | ARTERIAL HYPERTENSION | AMLODIPINE |
| 142 | CALCIUM CHANNEL BLOCKERS | ARTERIAL HYPERTENSION | VERAPAMIL |
| 143 | CALCIUM CHANNEL BLOCKERS | ATRIAL FIBRILLATION | DILTIAZEM |
| 144 | CALCIUM CHANNEL BLOCKERS | ELEVATED BLOOD PRESSURE | AMLODIPINE |
| 145 | CALCIUM CHANNEL BLOCKERS | ELEVATED BLOOD PRESSURE | AMLODIPINE BESILATE |
| 146 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL HYPERTENSION | AMLODIPINE |
| 147 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL HYPERTENSION | AMLODIPINE BESILATE |
| 148 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL HYPERTENSION | FELODIPINE |
| 149 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL PRIMARY<br>HYPERTENSION | AMLODIPINE |
| 150 | CALCIUM CHANNEL BLOCKERS | HIGH BLOOD PRESSURE | AMLODIPINE |
| 151 | CALCIUM CHANNEL BLOCKERS | HTN | AMLODIPINE |
| 152 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | AMLODIPINE |
| 153 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | AMLODIPINE BESILATE |
| 154 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | BARNIDIPINE<br>HYDROCHLORIDE |
| 155 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | DILTIAZEM |
| 156 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | DILTIAZEM HYDROCHLORIDE |
| 157 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | FELODIPINE |
| 158 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | NIFEDIPINE |
| 159 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | VERAPAMIL |
| 160 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION<br>(ESSENTIAL/PRIMARY) | VERAPAMIL HYDROCHLORIDE |
| 161 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION ESSENTIAL | FELODIPINE |
| 162 | CALCIUM CHANNEL BLOCKERS | HYPERTNESION | AMLODIPINE BESILATE |
| 163 | CALCIUM CHANNEL BLOCKERS | HYPTERTENSION | AMLODIPINE |
| 164 | CALCIUM CHANNEL BLOCKERS | PRESTUDY HYPERTENSION | AMLODIPINE |
| 165 | CALCIUM CHANNEL BLOCKERS | SECONDARY STROKE<br>PREVENTION | AMLODIPINE |
| 166 | CALCIUM CHANNEL BLOCKERS | SICK SINUS SYNDROME | VERAPAMIL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 167 | CALCIUM CHANNEL BLOCKERS | WORSENING OF<br>HYPERTENSION | AMLODIPINE |
| 168 | CARDIAC THERAPY | HYPERTENSION | UBIDECARENONE |
| 169 | DIURETICS | ARTERIAL HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 170 | DIURETICS | BENIGN ESSENTIAL<br>HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 171 | DIURETICS | BORDERLINE HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 172 | DIURETICS | DIURETIC | FUROSEMIDE |
| 173 | DIURETICS | ELEVATED BLOOD-PRESSURE<br>READING, WITHOUT<br>DIAGNOSIS OF HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 174 | DIURETICS | ESSENTIAL HYPERTENSION | FUROSEMIDE |
| 175 | DIURETICS | ESSENTIAL HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 176 | DIURETICS | HIGH BLOOD PRESSURE | HYDROCHLOROTHIAZIDE |
| 177 | DIURETICS | HYPERTENSION | AMILORIDE |
| 178 | DIURETICS | HYPERTENSION | BUMETANIDE |
| 179 | DIURETICS | HYPERTENSION | CHLORTALIDONE |
| 180 | DIURETICS | HYPERTENSION | DYAZIDE |
| 181 | DIURETICS | HYPERTENSION | FUROSEMIDE |
| 182 | DIURETICS | HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 183 | DIURETICS | HYPERTENSION | INDAPAMIDE |
| 184 | DIURETICS | HYPERTENSION | MODURETIC |
| 185 | DIURETICS | HYPERTENSION | SPIRONOLACTONE |
| 186 | DIURETICS | HYPERTENSION | TRIAMTERENE |
| 187 | DIURETICS | HYPERTENSION, BENIGN | HYDROCHLOROTHIAZIDE |
| 188 | DIURETICS | HYPERTENTION | HYDROCHLOROTHIAZIDE |
| 189 | DIURETICS | WORSENING HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 190 | LIPID MODIFYING AGENTS | HIGH BLOOD PRESSURE | PRAVASTATIN |
| 191 | LIPID MODIFYING AGENTS | HIGH BLOOD PRESSURE | PRAVASTATIN SODIUM |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| Diab | etes Mellitus (DIABETES) | | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | DIABETES MELLITUS TYPE II | LISINOPRIL |
| 2 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | TYPE 2 DIABETES | LISINOPRIL |
| 3 | ANTIHYPERTENSIVES | UNCONTROLLED DIABETES<br>MELLITUS 2 | CLONIDINE HYDROCHLORIDE |
| 4 | ANTIHYPERTENSIVES | UNCONTROLLED DIABETES<br>MELLITUS 2 | HYDRALAZINE<br>HYDROCHLORIDE |
| 5 | BETA BLOCKING AGENTS | TYPE 2 DIABETES | METOPROLOL TARTRATE |
| 6 | DRUGS USED IN DIABETES | BORDERLINE DIABETES | METFORMIN |
| 7 | DRUGS USED IN DIABETES | DIABETES | DULAGLUTIDE |
| 8 | DRUGS USED IN DIABETES | DIABETES | GLIBENCLAMIDE |
| 9 | DRUGS USED IN DIABETES | DIABETES | GLICLAZIDE |
| 10 | DRUGS USED IN DIABETES | DIABETES | GLIMEPIRIDE |
| 11 | DRUGS USED IN DIABETES | DIABETES | GLIPIZIDE |
| 12 | DRUGS USED IN DIABETES | DIABETES | HUMAN MIXTARD |
| 13 | DRUGS USED IN DIABETES | DIABETES | INSULIN |
| 14 | DRUGS USED IN DIABETES | DIABETES | INSULIN ASPART |
| 15 | DRUGS USED IN DIABETES | DIABETES | INSULIN DETEMIR |
| 16 | DRUGS USED IN DIABETES | DIABETES | INSULIN GLARGINE |
| 17 | DRUGS USED IN DIABETES | DIABETES | INSULIN HUMAN |
| 18 | DRUGS USED IN DIABETES | DIABETES | INSULIN LISPRO |
| 19 | DRUGS USED IN DIABETES | DIABETES | METAGLIP |
| 20 | DRUGS USED IN DIABETES | DIABETES | METFORMIN |
| 21 | DRUGS USED IN DIABETES | DIABETES | METFORMIN HYDROCHLORIDE |
| 22 | DRUGS USED IN DIABETES | DIABETES | PIOGLITAZONE |
| 23 | DRUGS USED IN DIABETES | DIABETES | PIOGLITAZONE<br>HYDROCHLORIDE |
| 24 | DRUGS USED IN DIABETES | DIABETES | SITAGLIPTIN |
| 25 | DRUGS USED IN DIABETES | DIABETES - TYPE I | INSULIN GLARGINE |
| 26 | DRUGS USED IN DIABETES | DIABETES - TYPE I | INSULIN LISPRO |
| 27 | DRUGS USED IN DIABETES | DIABETES 2 | GLICLAZIDE |
| 28 | DRUGS USED IN DIABETES | DIABETES II | METFORMIN |
| 29 | DRUGS USED IN DIABETES | DIABETES KETOACIDOSIS | INSULIN |
| 30 | DRUGS USED IN DIABETES | DIABETES MELL. TYPE 2 | INSULIN DETEMIR |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 31 | DRUGS USED IN DIABETES | DIABETES MELL. TYPE 2 | INSULIN LISPRO |
| 32 | DRUGS USED IN DIABETES | DIABETES MELL. TYPE 2 | METFORMIN |
| 33 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | EMPAGLIFLOZIN |
| 34 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | GLIBENCLAMIDE |
| 35 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | INSULIN DETEMIR |
| 36 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | INSULIN LISPRO |
| 37 | DRUGS USED IN DIABETES | DIABETES MELLITUS | DULAGLUTIDE |
| 38 | DRUGS USED IN DIABETES | DIABETES MELLITUS | EXENATIDE |
| 39 | DRUGS USED IN DIABETES | DIABETES MELLITUS | GLIPIZIDE |
| 40 | DRUGS USED IN DIABETES | DIABETES MELLITUS | HUMAN MIXTARD |
| 41 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN ASPART |
| 42 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN DETEMIR |
| 43 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN GLARGINE |
| 44 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN HUMAN |
| 45 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN LISPRO |
| 46 | DRUGS USED IN DIABETES | DIABETES MELLITUS | LIRAGLUTIDE |
| 47 | DRUGS USED IN DIABETES | DIABETES MELLITUS | METFORMIN |
| 48 | DRUGS USED IN DIABETES | DIABETES MELLITUS | METFORMIN HYDROCHLORIDE |
| 49 | DRUGS USED IN DIABETES | DIABETES MELLITUS | RISTFOR |
| 50 | DRUGS USED IN DIABETES | DIABETES MELLITUS | SITAGLIPTIN PHOSPHATE |
| 51 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYP II | INSULIN LISPRO |
| 52 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYP II | VELMETIA |
| 53 | DRUGS USED IN DIABETES | DIABETES MELLITUS 1 | INSULIN GLARGINE |
| 54 | DRUGS USED IN DIABETES | DIABETES MELLITUS 1 | INSULIN LISPRO |
| 55 | DRUGS USED IN DIABETES | DIABETES MELLITUS 11 | GLIPIZIDE |
| 56 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | CANAGLIFLOZIN |
| 57 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | DULAGLUTIDE |
| 58 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | EXENATIDE |
| 59 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | GLIBOMET |
| 60 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | GLIMEPIRIDE |
| 61 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | GLIPIZIDE |
| 62 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | HUMAN MIXTARD |
| 63 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | INSULIN ASPART |
| 64 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | INSULIN DETEMIR |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 65 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | INSULIN GLARGINE |
| 66 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | METFORMIN |
| 67 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | METFORMIN<br>HYDROCHLORIDE |
| 68 | DRUGS USED IN DIABETES | DIABETES MELLITUS II | GLIPIZIDE |
| 69 | DRUGS USED IN DIABETES | DIABETES MELLITUS II | METFORMIN |
| 70 | DRUGS USED IN DIABETES | DIABETES MELLITUS II | SITAGLIPTIN |
| 71 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYP 2 | METFORMIN |
| 72 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | GLIPIZIDE |
| 73 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | INSULIN GLARGINE |
| 74 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | INSULIN LISPRO |
| 75 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | METFORMIN |
| 76 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | METFORMIN<br>HYDROCHLORIDE |
| 77 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | SITAGLIPTIN PHOSPHATE |
| 78 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | CANAGLIFLOZIN<br>W/METFORMIN<br>HYDROCHLORIDE |
| 79 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | DULAGLUTIDE |
| 80 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | GLIPIZIDE |
| 81 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | HUMAN MIXTARD |
| 82 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN |
| 83 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN ASPART |
| 84 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN DETEMIR |
| 85 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN GLARGINE |
| 86 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN LISPRO |
| 87 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | METFORMIN |
| 88 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | METFORMIN HYDROCHLORIDE |
| 89 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | NATEGLINIDE |
| 90 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | SITAGLIPTIN PHOSPHATE |
| 91 | DRUGS USED IN DIABETES | DIABETES MELLITUS, TYPE II | METFORMIN HYDROCHLORIDE |
| 92 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | GLIPIZIDE |
| 93 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | HUMAN MIXTARD |
| 94 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN ASPART |
| 95 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN DETEMIR |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 96 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN GLARGINE |
| 97 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN LISPRO |
| 98 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | KOMBIGLYZE |
| 99 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | METFORMIN |
| 100 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | SITAGLIPTIN PHOSPHATE |
| 101 | DRUGS USED IN DIABETES | DIABETES TYPE II | METFORMIN |
| 102 | DRUGS USED IN DIABETES | DIABETES, TYPE 2 | GLIMEPIRIDE |
| 103 | DRUGS USED IN DIABETES | DIABETES, TYPE 2 | LIRAGLUTIDE |
| 104 | DRUGS USED IN DIABETES | DIABETES, TYPE 2 | PIOGLITAZONE |
| 105 | DRUGS USED IN DIABETES | DIABETIS | INSULIN GLARGINE |
| 106 | DRUGS USED IN DIABETES | DM2 | GLIPIZIDE |
| 107 | DRUGS USED IN DIABETES | DM2 | METFORMIN<br>HYDROCHLORIDE |
| 108 | DRUGS USED IN DIABETES | HYPERGLICEMIA | GLIPIZIDE |
| 109 | DRUGS USED IN DIABETES | HYPERGLYCEMIA | INSULIN HUMAN |
| 110 | DRUGS USED IN DIABETES | HYPERGLYCEMIA | METFORMIN |
| 111 | DRUGS USED IN DIABETES | HYPERGLYCEMIA | METFORMIN<br>HYDROCHLORIDE |
| 112 | DRUGS USED IN DIABETES | HYPERINSULINISM | METFORMIN |
| 113 | DRUGS USED IN DIABETES | HYPERTENSION | METFORMIN |
| 114 | DRUGS USED IN DIABETES | NONALCOHOLIC<br>STEATOHEPATITIS | METFORMIN |
| 115 | DRUGS USED IN DIABETES | TYPE 1 DIABETES | INSULIN DEGLUDEC |
| 116 | DRUGS USED IN DIABETES | TYPE 1 DIABETES MELLITUS | INSULIN ASPART |
| 117 | DRUGS USED IN DIABETES | TYPE 1 DIABETES MELLITUS | INSULIN GLARGINE |
| 118 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | GLICLAZIDE |
| 119 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | HUMAN MIXTARD |
| 120 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | INSULIN ASPART |
| 121 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | INSULIN GLARGINE |
| 122 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | INSULIN LISPRO |
| 123 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | METFORMIN |
| 124 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | METFORMIN<br>HYDROCHLORIDE |
| 125 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | SITAGLIPTIN PHOSPHATE |
| 126 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | GLIMEPIRIDE |
| | Medication Class (WHOATC2) Indication (CMINDC) | | WHOGEN |
|---|---|---|---|
| 127 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | HUMAN MIXTARD |
| 128 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | INSULIN HUMAN |
| 129 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | LIRAGLUTIDE |
| 130 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | METFORMIN<br>HYDROCHLORIDE |
| 131 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | PIOGLITAZONE |
| 132 | DRUGS USED IN DIABETES | TYPE II DIABETES | CANAGLIFLOZIN<br>W/METFORMIN<br>HYDROCHLORIDE |
| 133 | DRUGS USED IN DIABETES | TYPE II DIABETES | DAPAGLIFLOZIN<br>PROPANEDIOL<br>MONOHYDRATE W/METFO |
| 134 | DRUGS USED IN DIABETES | TYPE II DIABETES | GLIPIZIDE |
| 135 | DRUGS USED IN DIABETES | TYPE II DIABETES | INSULIN |
| 136 | DRUGS USED IN DIABETES | TYPE II DIABETES | INSULIN DETEMIR |
| 137 | DRUGS USED IN DIABETES | TYPE II DIABETES | INSULIN GLARGINE |
| 138 | DRUGS USED IN DIABETES | TYPE II DIABETES | LIRAGLUTIDE |
| 139 | DRUGS USED IN DIABETES | TYPE II DIABETES | METFORMIN |
| 140 | DRUGS USED IN DIABETES | TYPE II DIABETES | SITAGLIPTIN PHOSPHATE |
| 141 | DRUGS USED IN DIABETES | TYPE II DIABETES MELLITUS | EXENATIDE |
| 142 | DRUGS USED IN DIABETES | TYPE II DIABETES MELLITUS | METFORMIN |
| 143 | DRUGS USED IN DIABETES | TYPE II DIABETES MELLITUS | METFORMIN<br>HYDROCHLORIDE |
| 144 | DRUGS USED IN DIABETES | UNCONTROLLED DIABETES<br>MELLITUS 2 | INSULIN LISPRO |
| 145 | DRUGS USED IN DIABETES | UNCONTROLLED DIABETES<br>MELLITUS WITH<br>HYPERGLICEMIA | GLIPIZIDE |
| 146 | DRUGS USED IN DIABETES | UNCONTROLLED DIABETES<br>MELLITUS WITH<br>HYPERGLICEMIA | HUMAN MIXTARD |
| 147 | DRUGS USED IN DIABETES | UNCONTROLLED DM2 | INSULIN DETEMIR |
| 148 | UNSPECIFIED HERBAL AND<br>TRADITIONAL MEDICINE | HERBAL SUPPLEMENT | GLYCINE MAX EXTRACT |
| 149 | LIPID MODIFYING AGENTS | DIABETES MELLITUS TYPE II | PRAVASTATIN |

| | Medication Class (WHOATC2) Indication (CMINDC) | | WHOGEN |
|---|---|---|---|
| Card | liovascular (CARDDIS) | | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ACUTE MYOCARDIAL INFARCTION | IRBESARTAN |
| 2 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CARDIOMYOPATHY | LISINOPRIL |
| 3 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CARDIOMYOPATHY | RAMIPRIL |
| 4 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CONGESTIVE HEART FAILURE | LISINOPRIL |
| 5 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CORONARY ARTERY DISEASE | RAMIPRIL |
| 6 | BETA BLOCKING AGENTS | ACUTE MYOCARDIAL INFARCTION | BISOPROLOL FUMARATE |
| 7 | BETA BLOCKING AGENTS | ANTI-ARRHYTHMIC | SOTALOL |
| 8 | BETA BLOCKING AGENTS | ATHEROSCLEROTIC HEART<br>DISEASE OF NATIVE<br>CORONARY ARTERY<br>WITHOUT ANGINA PECTORIS | CARVEDILOL |
| 9 | BETA BLOCKING AGENTS | ATRIAL FIBRILATION | ATENOLOL |
| 10 | BETA BLOCKING AGENTS | ATRIAL FIBRILATION | METOPROLOL |
| 11 | BETA BLOCKING AGENTS | ATRIAL FIBRILLATION | METOPROLOL |
| 12 | BETA BLOCKING AGENTS | ATRIAL FIBRILLATION | METOPROLOL TARTRATE |
| 13 | BETA BLOCKING AGENTS | ATYPICAL CHEST PAIN | LABETALOL |
| 14 | BETA BLOCKING AGENTS | BRUGADA SYNDROME | BISOPROLOL |
| 15 | BETA BLOCKING AGENTS | CAD | METOPROLOL SUCCINATE |
| 16 | BETA BLOCKING AGENTS | CADRIOMYOPATHY | BISOPROLOL |
| 17 | BETA BLOCKING AGENTS | CARDIAC PACEMAKER INSITU | METOPROLOL |
| 18 | BETA BLOCKING AGENTS | CARDIAC PROPHYLAXIS | CARVEDILOL |
| 19 | BETA BLOCKING AGENTS | CARDIOMYOPATHY | CARVEDILOL |
| 20 | BETA BLOCKING AGENTS | CHEST TIGHTNESS | BISOPROLOL |
| 21 | BETA BLOCKING AGENTS | CONGESTIVE HEART FAILURE | ATENOLOL |
| 22 | BETA BLOCKING AGENTS | CONGESTIVE HEART FAILURE | CARVEDILOL |
| 23 | BETA BLOCKING AGENTS | CONTROLLED HYPERTENSION | TENORETIC |
| 24 | BETA BLOCKING AGENTS | CORONARY ARTERY DISEASE | METOPROLOL |
| 25 | BETA BLOCKING AGENTS | CORONARY ARTERY DISEASE | METOPROLOL SUCCINATE |
| 26 | BETA BLOCKING AGENTS | CORONARY ARTERY STENOSIS | METOPROLOL |
| 27 | BETA BLOCKING AGENTS | DYSRHYTHMIA | BISOPROLOL FUMARATE |
| 28 | BETA BLOCKING AGENTS | HEART FAILURE AND<br>HYPERTENSION | CARVEDILOL |
| 29 | BETA BLOCKING AGENTS | INTERMITTENT ARRHYTHMIA | BISOPROLOL |
| 30 | BETA BLOCKING AGENTS | MITRAL INSUFFICIENCY | BISOPROLOL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 31 | BETA BLOCKING AGENTS | PREVENTATIVE FOLLOWING<br>ACUTE MYCARDIAL<br>INFARCTION | BISOPROLOL |
| 32 | BETA BLOCKING AGENTS | SICK SINUS SYNDROME | METOPROLOL |
| 33 | BETA BLOCKING AGENTS | SUPRA VENTRICULAR<br>TACHYCARDIA | ATENOLOL |
| 34 | BETA BLOCKING AGENTS | SUPRAVENTRICULAR<br>TACHYCARDIA | ATENOLOL |
| 35 | BETA BLOCKING AGENTS | SUPRAVENTRICULAR<br>TACHYCARDIA | METOPROLOL |
| 36 | BETA BLOCKING AGENTS | TACHYCARDIA | ATENOLOL |
| 37 | CALCIUM CHANNEL BLOCKERS | CORONARY ARTERY DISEASE | AMLODIPINE |
| 38 | CALCIUM CHANNEL BLOCKERS | CORONARY ARTERY DISEASE | AMLODIPINE BESILATE |
| 39 | CALCIUM CHANNEL BLOCKERS | SUPRAVENTRICULAR<br>TACHYCARDIA | VERAPAMIL |
| 40 | CARDIAC THERAPY | ACUTE MYOCARDIAL INFARCTION | AMIODARONE<br>HYDROCHLORIDE |
| 41 | CARDIAC THERAPY | ACUTE MYOCARDIAL INFARCTION | ISOSORBIDE DINITRATE |
| 42 | CARDIAC THERAPY | ALLERGIC REACTION | EPINEPHRINE |
| 43 | CARDIAC THERAPY | ANGINA | GLYCERYL TRINITRATE |
| 44 | CARDIAC THERAPY | ANGINA PECTORIS | RANOLAZINE |
| 45 | CARDIAC THERAPY | ANGIOGRAM/STENT | ADENOSINE |
| 46 | CARDIAC THERAPY | ANGIONEUROTIC EDEMA | EPINEPHRINE |
| 47 | CARDIAC THERAPY | ANTIARRHYTHMIC AGENT | FLECAINIDE ACETATE |
| 48 | CARDIAC THERAPY | ATRIAL FIBRILLATION | DIGOXIN |
| 49 | CARDIAC THERAPY | ATRIAL FIBRILLATION | FLECAINIDE ACETATE |
| 50 | CARDIAC THERAPY | ATYPICAL CHEST PAIN | GLYCERYL TRINITRATE |
| 51 | CARDIAC THERAPY | CAD | UBIDECARENONE |
| 52 | CARDIAC THERAPY | CARDIOMYOPATHY | ISOSORBIDE DINITRATE |
| 53 | CARDIAC THERAPY | CARDIOVASCULAR DISEASE<br>PROPHYLAXIS | UBIDECARENONE |
| 54 | CARDIAC THERAPY | CHEST PAIN | GLYCERYL TRINITRATE |
| 55 | CARDIAC THERAPY | CHEST PAINS | GLYCERYL TRINITRATE |
| 56 | CARDIAC THERAPY | CHESTPAIN | GLYCERYL TRINITRATE |
| 57 | CARDIAC THERAPY | CORONARY ARTERY DISEASE | GLYCERYL TRINITRATE |
| 58 | CARDIAC THERAPY | CORONARY ARTERY DISEASE | ISOSORBIDE MONONITRATE |
| 59 | CARDIAC THERAPY | HYPERLIPIDEMIA | ISOSORBIDE MONONITRATE |
| 60 | CARDIAC THERAPY | NSTEMI | ISOSORBIDE DINITRATE |
| 61 | CARDIAC THERAPY | PERIOP STRESS TEST | REGADENOSON |
| 62 | CARDIAC THERAPY | PROPHYLAXIS | GLYCERYL TRINITRATE |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 63 | CARDIAC THERAPY | PROPHYLAXIS FOR CARDIAC HEALTH | UBIDECARENONE |
| 64 | CARDIAC THERAPY | SUPRAVENTRICULAR<br>TACHYCARDIA | ADENOSINE |
| 65 | CARDIAC THERAPY | UNCONTROLLED DIABETES<br>MELLITUS 2 | AMIODARONE<br>HYDROCHLORIDE |
| 66 | CARDIAC THERAPY | UNCONTROLLED DIABETES MELLITUS 2 | GLYCERYL TRINITRATE |
| 67 | DIURETICS | ACUTE RESPIRATORY<br>FAILURE | FUROSEMIDE |
| 68 | DIURETICS | AORTIC VALVE<br>REPLACEMENT | FUROSEMIDE |
| 69 | DIURETICS | CHF | BUMETANIDE |
| 70 | DIURETICS | CHF | HYDROCHLOROTHIAZIDE |
| 71 | DIURETICS | CHF | METOLAZONE |
| 72 | DIURETICS | CONGESTIVE HEART FAILURE | BUMETANIDE |
| 73 | DIURETICS | CONGESTIVE HEART FAILURE | FUROSEMIDE |
| 74 | DIURETICS | CONGESTIVE HEART FAILURE | HYDROCHLOROTHIAZIDE |
| 75 | DIURETICS | CONGESTIVE HEART FAILURE | METOLAZONE |
| 76 | DIURETICS | CONGESTIVE HEART FAILURE | SPIRONOLACTONE |
| 77 | DIURETICS | CORONARY ARTERY DISEASE | HYDROCHLOROTHIAZIDE |
| 78 | DIURETICS | CORONARY ARTERY DISEASE. | FUROSEMIDE |
| 79 | DIURETICS | ELEVATION OF BLOOD<br>PRESSURE | FUROSEMIDE |
| 80 | DIURETICS | MITRAL INSUFFICIENCY | TORASEMIDE |
| 81 | DIURETICS | TRANSGENGER | SPIRONOLACTONE |
| 82 | LIPID MODIFYING AGENTS | ACUTE MYOCARDIAL INFARCTION | ATORVASTATIN CALCIUM |
| 83 | LIPID MODIFYING AGENTS | ACUTE MYOCARDIAL INFARCTION | OMEGA-3 TRIGLYCERIDES |
| 84 | LIPID MODIFYING AGENTS | ATHEROSCLEROTIC HEART<br>DISEASE OF NATIVE<br>CORONARY ARTERY<br>WITHOUT ANGINA PECTORIS | SIMVASTATIN |
| 85 | LIPID MODIFYING AGENTS | BASILAR ARTERY THROMBUS | ATORVASTATIN CALCIUM |
| 86 | LIPID MODIFYING AGENTS | CAD | PRAVASTATIN SODIUM |
| 87 | LIPID MODIFYING AGENTS | CAD | ROSUVASTATIN CALCIUM |
| 88 | LIPID MODIFYING AGENTS | CARDIAC PROPHYLAXIS | ATORVASTATIN |
| 89 | LIPID MODIFYING AGENTS | CARDIAC PROPHYLAXIS | FISH OIL |
| 90 | LIPID MODIFYING AGENTS | CARDIOVASCULAR<br>PROPHYLAXIS | ATORVASTATIN CALCIUM |
| 91 | LIPID MODIFYING AGENTS | CHEST TIGHTNESS | ATORVASTATIN |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| Нуре | Hyperlipidemia (HLIPDEM) | | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTRIGLYCERIDEMIA | LISINOPRIL |
| 2 | ANTIHYPERTENSIVES | HYPERCHOLESTEROLEMIA | DOXAZOSIN MESILATE |
| 3 | CARDIAC THERAPY | HYPERCHOLESTEROLEMIA | UBIDECARENONE |
| 4 | LIPID MODIFYING AGENTS | ABNORMAL LIPIDS | ATORVASTATIN |
| 5 | LIPID MODIFYING AGENTS | CARDIAC PROPHYLAXIS | ROSUVASTATIN |
| 6 | LIPID MODIFYING AGENTS | CHOLESTEROL | ROSUVASTATIN |
| 7 | LIPID MODIFYING AGENTS | CHOLESTEROL | ROSUVASTATIN CALCIUM |
| 8 | LIPID MODIFYING AGENTS | CHOLESTEROLEAMIA | ATORVASTATIN |
| 9 | LIPID MODIFYING AGENTS | CHOLESTERORL | ROSUVASTATIN CALCIUM |
| 10 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | ATORVASTATIN |
| 11 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | EZETIMIBE |
| 12 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | FENOFIBRATE |
| 13 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | ROSUVASTATIN CALCIUM |
| 14 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE PROPHYLAXIS | ATORVASTATIN |
| 15 | LIPID MODIFYING AGENTS | DIET SUPPLEMENT | FISH OIL |
| 16 | LIPID MODIFYING AGENTS | DIETARY SUPPLEMENT | FISH OIL |
| 17 | LIPID MODIFYING AGENTS | DIETARY SUPPLEMENTS | FISH OIL |
| 18 | LIPID MODIFYING AGENTS | DYSLIPEDEMIA | ROSUVASTATIN CALCIUM |
| 19 | LIPID MODIFYING AGENTS | DYSLIPIDAEMIA | ATORVASTATIN |
| 20 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | ATORVASTATIN |
| 21 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | FENOFIBRATE |
| 22 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | FISH OIL |
| 23 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | GEMFIBROZIL |
| 24 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | PRAVASTATIN |
| 25 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | ROSUVASTATIN |
| 26 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA, WORSENING | ROSUVASTATIN |
| 27 | LIPID MODIFYING AGENTS | DYSLIPIDERMIA | PRAVASTATIN |
| 28 | LIPID MODIFYING AGENTS | ELEVATED CHOLESTEROL | SIMVASTATIN |
| 29 | LIPID MODIFYING AGENTS | ELEVATED LIPIDS | ATORVASTATIN |
| 30 | LIPID MODIFYING AGENTS | ELEVATED LIPIDS | ATORVASTATIN CALCIUM |
| 31 | LIPID MODIFYING AGENTS | ELEVATED TRIGLYCERIDES | FISH OIL |
| 32 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | ATORVASTATIN |

| | Medication Class (WHOATC2) Indication (CMINDC) | | WHOGEN |
|---|---|---|---|
| 33 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | ATORVASTATIN CALCIUM |
| 34 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | GEMFIBROZIL |
| 35 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | LOVASTATIN |
| 36 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | PRAVASTATIN |
| 37 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | ROSUVASTATIN CALCIUM |
| 38 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | SIMVASTATIN |
| 39 | LIPID MODIFYING AGENTS | HIGH CHOLESTROL | ATORVASTATIN |
| 40 | LIPID MODIFYING AGENTS | HIGH PLASMA LIPIDS | ATORVASTATIN |
| 41 | LIPID MODIFYING AGENTS | HIGH TRIGLYCERIDES | FENOFIBRATE |
| 42 | LIPID MODIFYING AGENTS | HIGH TRIGLYCERIDES AND<br>HYPERCHOLESTEROLEMIA | ATORVASTATIN |
| 43 | LIPID MODIFYING AGENTS | HIPERCOLESTEROLEMIA | ATORVASTATIN |
| 44 | LIPID MODIFYING AGENTS | HIPERCOLESTEROLEMIA | ATORVASTATIN CALCIUM |
| 45 | LIPID MODIFYING AGENTS | HIPERCOLESTEROLEMIA | SIMVASTATIN |
| 46 | LIPID MODIFYING AGENTS | HYERLIPIDEMIA | OMEGA-3-ACID ETHYL ESTER |
| 47 | LIPID MODIFYING AGENTS | HYPERCHOLESTERIMIA | FENOFIBRATE |
| 48 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINAEMIA | ATORVASTATIN |
| 49 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINAEMIA | PRAVASTATIN |
| 50 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINEMIA | PRAVASTATIN |
| 51 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINEMIA | SIMVASTATIN |
| 52 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROL | PRAVASTATIN |
| 53 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | ATORVASTATIN |
| 54 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | PRAVASTATIN |
| 55 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | ROSUVASTATIN |
| 56 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | SIMVASTATIN |
| 57 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ATORVASTATIN |
| 58 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ATORVASTATIN CALCIUM |
| 59 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | EZETIMIBE |
| 60 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | FENOFIBRATE |
| 61 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | FISH OIL |
| 62 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | LOVASTATIN |
| 63 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | PITAVASTATIN CALCIUM |
| 64 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | PRAVASTATIN |
| 65 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | PRAVASTATIN SODIUM |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 66 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ROSUVASTATIN |
| 67 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ROSUVASTATIN CALCIUM |
| 68 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | SIMVASTATIN |
| 69 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA<br>(PURE) AND MIXED<br>HYPERLIPIDEMIA | ROSUVASTATIN CALCIUM |
| 70 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLMIA | PRAVASTATIN SODIUM |
| 71 | LIPID MODIFYING AGENTS | HYPERCHOLESTROLEMIA | ATORVASTATIN |
| 72 | LIPID MODIFYING AGENTS | HYPERCHOLESTROLEMIA | ATORVASTATIN CALCIUM |
| 73 | LIPID MODIFYING AGENTS | HYPERCHOLESTROLEMIA | FENOFIBRATE |
| 74 | LIPID MODIFYING AGENTS | HYPERCHOLSTEROAEMIA | ATORVASTATIN CALCIUM |
| 75 | LIPID MODIFYING AGENTS | HYPERCOLESTEROLEMIA | SIMVASTATIN |
| 76 | LIPID MODIFYING AGENTS | HYPERLIDEMIA | ROSUVASTATIN CALCIUM |
| 77 | LIPID MODIFYING AGENTS | HYPERLIDIPEMIA | ATORVASTATIN |
| 78 | LIPID MODIFYING AGENTS | HYPERLIPDEMIA | ROSUVASTATIN CALCIUM |
| 79 | LIPID MODIFYING AGENTS | HYPERLIPEDMIA-MIXED | ATORVASTATIN |
| 80 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | ATORVASTATIN |
| 81 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | FENOFIBRATE |
| 82 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | PRAVASTATIN |
| 83 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | PRAVASTATIN SODIUM |
| 84 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | ROSUVASTATIN |
| 85 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | ROSUVASTATIN CALCIUM |
| 86 | LIPID MODIFYING AGENTS | HYPERLIPIDEMA | ATORVASTATIN |
| 87 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ATORVASTATIN |
| 88 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ATORVASTATIN CALCIUM |
| 89 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | COLESEVELAM<br>HYDROCHLORIDE |
| 90 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | EICOSAPENTAENOIC ACID<br>ETHYL ESTER |
| 91 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | EZETIMIBE |
| 92 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | FENOFIBRATE |
| 93 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | FENOFIBRIC ACID |
| 94 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | FISH OIL |
| 95 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | GEMFIBROZIL |
| 96 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | LOVASTATIN |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 97 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | OMEGA-3-ACID ETHYL ESTER |
| 98 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | PELAGO |
| 99 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | PRAVASTATIN |
| 100 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | PRAVASTATIN SODIUM |
| 101 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ROSUVASTATIN |
| 102 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ROSUVASTATIN CALCIUM |
| 103 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | SIMVASTATIN |
| 104 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA<br>PREVENTION | ROSUVASTATIN CALCIUM |
| 105 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA, | PRAVASTATIN |
| 106 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA, MIXED | ATORVASTATIN CALCIUM |
| 107 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA, MIXED | FENOFIBRATE |
| 108 | LIPID MODIFYING AGENTS | HYPERTENSION | ATORVASTATIN |
| 109 | LIPID MODIFYING AGENTS | HYPERTENSION | PRAVASTATIN |
| 110 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERDEMIA | ATORVASTATIN |
| 111 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | ATORVASTATIN CALCIUM |
| 112 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FENOFIBRATE |
| 113 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FENOFIBRIC ACID |
| 114 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FIBRATES |
| 115 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FISH OIL |
| 116 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | OMEGA-3 TRIGLYCERIDES |
| 117 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | PRAVASTATIN |
| 118 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA,HY<br>PERCHOLESTEROLEMIA | ATORVASTATIN |
| 119 | LIPID MODIFYING AGENTS | HYPERTRIGLYERIDEMIA | GEMFIBROZIL |
| 120 | LIPID MODIFYING AGENTS | HYPERTRYGLYCERIDEMIA | PRAVASTATIN |
| 121 | LIPID MODIFYING AGENTS | INDICATION HYPERLIPIDEMIA | FENOFIBRATE |
| 122 | LIPID MODIFYING AGENTS | IRRITABLE BOWEL<br>SYNDROME | FISH OIL |
| 123 | LIPID MODIFYING AGENTS | ISCHEMIC HEART DISEASE | ROSUVASTATIN CALCIUM |
| 124 | LIPID MODIFYING AGENTS | LDL-CHOLESTEROL GRADE 3<br>ELEVATION | ROSUVASTATIN |
| 125 | LIPID MODIFYING AGENTS | MIXED DYSLIPIDEMIA | FENOFIBRATE |
| 126 | LIPID MODIFYING AGENTS | MIXED DYSLIPIDEMIA | ROSUVASTATIN CALCIUM |
| 127 | LIPID MODIFYING AGENTS | MIXED HYPERLIPDEMIA | ATORVASTATIN |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 128 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | ATORVASTATIN |
| 129 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | FENOFIBRATE |
| 130 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | GEMFIBROZIL |
| 131 | LIPID MODIFYING AGENTS | NUTRITION SUPPLEMENT | FISH OIL |
| 132 | LIPID MODIFYING AGENTS | NUTRITIONAL SUPPLEMENT | FISH OIL |
| 133 | LIPID MODIFYING AGENTS | NUTRITIONAL SUPPLEMENT | OMEGA-3 FATTY ACIDS |
| 134 | LIPID MODIFYING AGENTS | PREVENTATIVE FOLLOWING<br>ACUTE MYCARDIAL<br>INFARCTION | ATORVASTATIN |
| 135 | LIPID MODIFYING AGENTS | PREVENTION FOR<br>HYPERCHOLESTEROLEMIA | OMEGA-3 FATTY ACIDS |
| 136 | LIPID MODIFYING AGENTS | PREVENTIVE | FISH OIL W/LINUM<br>USITATISSIMUM SEED OIL |
| 137 | LIPID MODIFYING AGENTS | PROPHYLAXIS | FISH OIL |
| 138 | LIPID MODIFYING AGENTS | PURE<br>HYPERCHOLESTEROLEMIA | ATORVASTATIN |
| 139 | LIPID MODIFYING AGENTS | SECONDARY STROKE<br>PREVENTION | ATORVASTATIN |
| 140 | LIPID MODIFYING AGENTS | STROKE PROPHYLAXIS | ATORVASTATIN |
| 141 | LIPID MODIFYING AGENTS | SUPPLEMENT | FISH OIL |
| 142 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA 3 6 9 |
| 143 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA-3 FATTY ACIDS |
| 144 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA-3 FATTY ACIDS<br>W/OMEGA-6 FATTY ACIDS |
| 145 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA-3-ACID ETHYL ESTER |
| 146 | LIPID MODIFYING AGENTS | SUPPLEMENT/HYPERLIPIDEMIA | FISH OIL |
| 147 | LIPID MODIFYING AGENTS | SUPPLEMENTAL USE | FISH OIL |
| 148 | LIPID MODIFYING AGENTS | SUPPLEMETN | FISH OIL |
| 149 | LIPID MODIFYING AGENTS | UNCONTROLLED DIABETES<br>MELLITUS 2 | ATORVASTATIN |
| 150 | LIPID MODIFYING AGENTS | WORSENING HYPERLIPIDEMIA | ATORVASTATIN |
| 151 | LIPID MODIFYING AGENTS | WORSENING OF<br>HYPERLIPIDEMIA | FISH OIL |
| 152 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | NICOTINIC ACID |
| 153 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | NICOTINIC ACID |
| 154 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | NICOTINIC ACID |
| 155 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | NICOTINIC ACID |

# **Appendix 5.** Hepatic Events

An adverse event record will be flagged as a hepatic event if its MedDRA PT included in the pre-specified PT list, which includes all PTs from the broad search of the following 15 SMQs under MedDRA 19.1 provided by Gilead DSPH and reviewed by Gilead medical monitors.

| | SMQ Source |
|---|---|
| | Biliary neoplasms benign (incl cysts and polyps) (SMQ) |
| | Biliary malignant tumours (SMQ) |
| | Biliary tumours of unspecified malignancy (SMQ) |
| | Biliary system related investigations, signs and symptoms (SMQ) |
| | Biliary tract disorders (SMQ) |
| | Gallbladder related disorders (SMQ) |
| | Gallstone related disorders (SMQ) |
| Hepatic Events (HEP) | Cholestasis and jaundice of hepatic origin (SMQ) |
| | Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ) |
| | Hepatitis, non-infectious (SMQ) |
| | Liver neoplasms, benign (incl cysts and polyps) (SMQ) |
| | Liver malignant tumours (SMQ) |
| | Liver tumours of unspecified malignancy (SMQ) |
| | Liver related investigations, signs and symptoms (SMQ) |
| | Liver-related coagulation and bleeding disturbances (SMQ) |

# **Appendix 6. Programming Specification**

- 1) AGE calculated as follows:
  - a) AGE (years) is calculated from the number of days between the date of birth (DOB) and Day 1 (first dose date),
  - b) Use the SAS INTCK function to determine the number of "1st-of-month days" (eg, January 1st, February 1st, March 1st) between DOB and Day 1 (inclusive),
  - c) Divide the result in (b) by 12,
  - d) AGE = the integer of the result in (c),
  - e) If the DOB and Day 1 have the month in common and the birthday is later in the month than the date of Study Day 1, then subtract one from the AGE result above.

For subjects randomized and never dosed with study drug, age will be calculated from the date of randomization.

- 2) All screened subjects refer to all subjects who are screened (ie, with nonmissing screening date) and have a screening number. For summaries, the same subject is counted only once. DOB and other demographic information such as sex, race, ethnicity, country, and initials will be used to identify unique screened subjects.
- 3) Screen failure subjects are the subjects who are screened and answered "No" for any inclusion criteria or "Yes" for any exclusion criteria regardless of which version of protocol the subject was consent to.
- 4) Subjects in the randomized analysis set are defined as subjects randomized into the study. IXRSRAND is the source to determine whether the subject is randomized (ie, subject with nonmissing RGMNDTN in the IXRSRAND dataset) and confirmed by the eCRF ENROLL dataset (ie, ENROLLYN = "Yes" in ENROLL dataset).
- 5) Randomized treatment (ie, TRT01P in ADSL) are derived from IXRSRAND, while actual treatment received (ie, TRT01A in ADSL) is assigned as the randomized treatment if subject took at least 1 dose of study drug and assigned as blank if subject never dosed.
- 6) Enrollment by Stratum: using actual HIV-1 RNA or CD4+ cell count screening value, the last screening value (with visitnum < 0) prior to randomization date and time.
- 7) In disposition table, the reasons for premature discontinuation are displayed in the order as they appear on the eCRF.

8) Body mass index (BMI) and Body Surface Area (BSA)

BMI and BSA will be calculated only at baseline as follows:

- BMI = (weight [kg])/ (height [meters]<sup>2</sup>)
- BSA  $(m^2)$  = SQRT( [Height(cm) x Weight(kg) ]/ 3600 )

Baseline height and weight will be used for this calculation.

- 9) SAS codes for the treatment comparison for demographics and baseline characteristics tables.
  - a) CMH test for nominal variable (Y), the p-value from general association test should be used for nominal variable:

```
proc freq order=adsl;
  tables trtgrp * Y /cmh /*general association test*/
run;
```

b) CMH test for ordinal variable (Y), the p-value from row mean score test should be used for ordinal variable:

```
proc freq order=adsl;
  tables trtgrp * Y / cmh2 ; /*row mean score test*/
run;
```

c) Wilcoxon rank sum test for continuous variable (Y), the p-value from the normal approximation two-sided test should be used for continuous variable:

```
proc npar1way wilcoxon data=adsl;
  class trtgrp;
  var Y;
run;
```

10) Please note, "Not Permitted", "Unknown", or missing categories will be excluded for percentage calculation and also excluded for p value generation for categorical data analysis (eg, CMH test or Fisher exact test). Except for Mode of infection (HIV Risk Factors), where "Unknown" will be included for percentage calculation, since a subject may fit more than 1 HIV risk factors, therefore percentage may add to more than 100% and no p-value will be generated.

Subjects with Race = "Not Permitted" will also be excluded to define Race subgroup (ie, black vs. nonblack) for efficacy subgroup analysis.

11) SAS code for the treatment comparison for duration of exposure. The p-value from log rank test should be used.

```
proc lifetest data=ADSL method=km;
  time TRTDURD*ESDD(0); /*Derive ESDD from COMT01FL, where ESDD = 0
  indicates censored observation (ie, subject is still on study drug)*/
  Strata TRT01AN;
  label TRTDURD = "Duration of Exposure (Days)";
run;
```

- 12) Last Dose Date and Last Study Date
  - a) Last Dose Date (ie, TRTEDTC, TRTEDT, TR01EDT or TR01EDTC) in ADSL was defined in Section 3.8.1.

For subjects with a partial last dosing date (ie, month and year of last dose are known), the latest of the dispensing dates of study drug bottles, study drug start dates and end dates, and the imputed last dose date [day imputed as 15] will be used as the final imputed last dose date. However if dispensing date's month is after last dose date's month, data query is needed.

If subject died and the death date is complete (ie, not partial date) and before the imputed last dose date, the complete death date should be used as the imputed last dose date.

Last dose date is not defined for subjects still on study drug in SAP. However, for the calculation of the duration of exposure to study drug, the data cut date will be used to impute the last dose date for subjects who have not permanently discontinued study drug at the time of the data cut date.

For Week 48 interim analysis, 05/11/2017 will be the data cut date for subjects with Week 48 visits on or prior to 05/11/2017, subjects missing week 48 visits while on study drug, or subjects prematurely discontinued study drug. For subjects with Week 48 visit after 05/11/2017, the last subject's week 48 visit will be used as the data cut date as appropriate.

b) Last Study Date is the latest of the study drug start dates and end dates, the clinic visit dates, and the laboratory visit dates, including the 30-day follow-up visit date, for subjects who prematurely discontinued study or who completed study according to the Study Completion eCRF. If study drug start dates or end date is partially missing (ie, only year and month are known), the day will be imputed as 15 for the purpose of this analysis.

If subject died and the death date is complete (ie, not partial date) and before the imputed last study date, the complete death date should be used as the imputed last study date. Last study date is not defined for subjects still on study in SAP. However, for programing purposes, the latest of data cut date, the clinic visit dates, and the laboratory visit dates, including the 30-day follow-up visit date, will be used to impute the last study date for subjects still on study.

# 13) Toxicity Grades:

- a) For toxicity grade summaries, include all post-baseline graded results up to 30 days after the last dose of study drug, not just those used in by-visit summaries.
- b) For glucose grading, as specified in SAP Section 7.2.2.1, the treatment-emergent flag cannot be determined for nonfasting glucose (including glucose results without a known fasting status). As a result, these records will be excluded from the "Maximum Treatment-emergent Toxicity Grade" summary in the "Treatment-emergent Laboratory Abnormalities" or "Treatment-emergent Grade 3 or 4 Laboratory Abnormalities" summary tables. In addition, fasting glucose and nonfasting glucose will be listed as two separate laboratory tests in the "Laboratory Abnormalities" and "Grade 3 or 4 Laboratory Abnormalities" listings. Only a maximum postbaseline toxicity flag will be displayed and the treatment-emergent flag will not be displayed for nonfasting glucose as the treatment-emergent flag cannot be determined for nonfasting glucose.

#### 14) Efficacy analyses:

a) For categorical efficacy response (eg, Subjects with HIV-1 RNA < 50 copies/mL as determined by US FDA-defined snapshot algorithm, M=F, or M=E Analyses): the proportion difference between two treatment groups and its 95.002% or 95% CIs are calculated based on the MH proportion adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US) (see SAP Section 6.1.4 for details). To test superiority, the p-value from 2-sided CMH test (ie, general association test) stratified by baseline HIV-1 RNA stratum and region stratum should be used, where *brnac* is the baseline HIV-1 RNA stratum, *region* is the region stratum, *trtgrp* is the treatment, and *response* is the categorical efficacy response. The following SAS code will be used to compute cell counts and p-value.

```
proc freq data=adeff;
   tables brnac*region*trtgrp*response/cmh; /*p value from general
   association*/
run;
```

b) Homogeneity test: Homogeneity Test of Treatment Effect Across Region in HIV-1 RNA < 50 copies/mL at Week 48 (Snapshot Algorithm). For each region, the odds ratio and its 95% CI are calculated from the CMH test. For overall, the odds ratio and its 95% CI are calculated based on the common odds ratio estimate from the CMH test. The p-value for the homogeneity test is based on the Breslow-Day test of the interaction between region and treatment group as follows.

```
proc freq data=adeff;
   tables region2*trtgrp*response/all; /*p value from Breslow Day test*/
run:
```

- c) Subgroup analyses
  - i) For the subgroups of age, sex, race, baseline CD4+ cell count, and study drug adherence, the proportion difference between two treatment groups and its 95% CIs are calculated based on the MH proportion adjusted by **baseline HIV-1 RNA stratum and region stratum** (see Section 6.1.4 for details). For example, for the age subgroup, the following SAS code will be used to compute cell counts.

```
proc sort data=adeff;
   by agegrp brnac region;
proc freq data=adeff;
   by agegrp;
   tables brnac*region*trtgrp*response/cmh;
run;
```

ii) For the baseline HIV-1 RNA subgroup, the proportion difference between two treatment groups and its 95% CIs are calculated based on the MH proportion adjusted by **region stratum** only. The following SAS code will be used to compute the cell counts.

```
proc sort data=adeff;
   by brnac region;
proc freq data=adeff;
   by brnac;
   tables region*trtgrp*response/ cmh;
run;
```

iii) For the region subgroup, the proportion difference between two treatment groups and its 95% CIs are calculated based on the MH proportion adjusted by **baseline HIV-1 RNA stratum** only. The following SAS code will be used to compute the cell counts.

```
proc sort data=adeff;
  by region brnac;
proc freq data=adeff;
  by region;
  tables brnac*trtgrp*response/ cmh;
run;
```

- d) Homogeneity test: Homogeneity Test of Treatment Effect between Subgroups in HIV-1 RNA < 50 copies/mL at Week 48 (Snapshot Algorithm)
  - i) For the subgroups of age, sex, race, baseline CD4+ cell count, and study drug adherence, the odds ratio and the associated 95% CIs are estimated for the response variable (response; coded as 1 for success and 0 for non-success) using a logistic regression model including treatment (trtgrp; coded as 1 for active [ie, B/F/TAF] and 2 for control), baseline HIV-1 RNA stratum (brnac; coded as 1 for < 100,000 copies/mL and 2 for >= 100,000 copies/mL), region stratum (region; coded as 1 for "US" and 2 for "Ex-US"), subgroup factor (coded as 1 for the first subgroup and 2 for the second subgroup), and treatment by subgroup factor. For example, for the age subgroup (agegrp; coded as 1 for < 50 and 2 for >= 50), the following SAS code will be used to generate the Odds Ratio and its 95% CI within the subgroup:

Note: For the following code, it is assumed that none of the variables have any formats applied to them. If they do, they must be removed before calling the code.

```
proc genmod data=data descending; /*model for success*/
   class trtgrp brnac region agegrp;
   model response = trtgrp brnac region agegrp trtgrp*agegrp/dist=bin
   link=logit lrci;
   estimate 'Group 1' trtgrp 1 -1 trtgrp*agegrp 1 0 -1 0/exp;
   estimate 'Group 2' trtgrp 1 -1 trtgrp*agegrp 0 1 0 -1/exp;
run;
```

ii) For the baseline HIV-1 RNA subgroups, the odds ratio and the associated 95% CIs are estimated using a logistic regression model including treatment, region stratum, subgroup factor, and treatment by subgroup factor. The following SAS code will be used to generate the Odds Ratio and its 95% CI within the subgroup (the same formats as described in (a) above are assumed):

```
proc genmod data=data descending;
  class trtgrp region brnac;
  model response = trtgrp region brnac trtgrp* brnac/dist=bin link=logit lrci;
  estimate 'Group 1' trtgrp 1 -1 trtgrp*brnac 1 0 -1 0/exp;
  estimate 'Group 2' trtgrp 1 -1 trtgrp*brnac 0 1 0 -1/exp;
run;
```

iii) For the region subgroups, the odds ratio and the associated 95% CIs are estimated using a logistic regression model including treatment, baseline HIV-1 RNA stratum, subgroup factor, and treatment by subgroup factor. The following SAS code will be used to generate the Odds Ratio and its 95% CI within the subgroup (the same formats as described in (a) above are assumed):

```
proc genmod data=data descending;
   class trtgrp brnac region;
   model response = trtgrp brnac region trtgrp*region/dist=bin link=logit lrci;
   estimate 'Group 1' trtgrp 1 -1 trtgrp*region 1 0 -1 0/exp;
   estimate 'Group 2' trtgrp 1 -1 trtgrp*region 0 1 0 -1/exp;
run;
```

- if  $n_{1h}$  or  $n_{2h} > 1$  the denominator  $n_{1h} 1$  or  $n_{2h} 1$  was calculated as indicated in the formula:
- if  $n_{1h}$  or  $n_{2h} = 1$ , the corresponding  $n_{1h}$  or  $n_{2h}$  will be adjusted to 2, then corresponding denominator  $[(n_{1h} 1) \text{ or } (n_{2h} 1)]$  is 1;
- if  $n_{1h}$  or  $n_{2h} = 0$  but not both  $n_{1h}$  and  $n_{2h} = 0$  then not calculable;
- if both  $n_{1h}$  and  $n_{2h} = 0$  then the corresponding stratum will be ignored, will not be included in the calculation, thus the proportion difference and 95% CI are still calculable.

If the sample size in a subgroup is too small to calculate the proportion difference between 2 treatment groups and its 95% CI based on the stratum-adjusted MH proportion, then a 95% CI based on the normal approximation will be used. For example, if the stratum-adjusted MH proportion cannot be calculated for sex = "Female" subgroup, the following code will be used to calculate the proportion difference and 95% CI based on the normal approximation, ie, *riskdiff* option in *tables* statement will provide the proportion difference and 95% CI estimations.

```
proc freq data = adeff;
   where sex = "F";
   tables trtgrp*response/ riskdiff(CL=(WALD));
run;
```

e) ANOVA model for continuous efficacy variable (eg, CD4+): The differences in changes from baseline in CD4+ cell count between treatment groups and the associated 95% CI will be constructed using an ANOVA, including baseline HIV-1 RNA stratum, region stratum, and treatment as fixed effects in the model.

```
proc glm data=adeff;
   class brnac region trtgrp;
   model CD4=brnac region trtgrp;
   lsmeans trtgrp /alpha=0.05 cl pdiff;
run;
```

f) Listing for US FDA-defined snapshot outcome:

In addition to flagging the values of HIV-1 RNA < 50 or  $\ge 50$  copies/mL for virologic outcomes, flag the last available HIV-1 RNA value while on treatment for the following categories:

- i) HIV-1 RNA  $\geq$  50 copies/mL Discontinued Study Drug Due to Other Reasons and Last Available HIV-1 RNA  $\geq$  50 copies/mL
- ii) No virologic Data Discontinued Study Drug Due to Other Reasons and Last Available HIV-1 RNA < 50 copies/mL

#### 15) TEAE

# **Events with Missing Onset Day and/or Month**

An AE is treatment emergent if the following 3 criteria are met:

- 1) The month and year (or year) of onset date is the same as or after the month and year (or year) of the first dose of study drug, and
- 2) The month and year (or year) of the onset date is the same as or before the month and year (or year) of the 30th day after the date of the last dose of study drug, and
- 3) End date is as follows:
  - a) The (complete) end date is on or after the first dose date, or
  - b) The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of study drug, or
  - c) End date is completely missing

#### **Events with Completely Missing Onset Date**

An AE with a completely missing onset date is defined as TEAE if end date meets any of the criteria specified in 3) above.

#### 16) Graded Laboratory Abnormalities Summary

The following labels will be used for treatment-emergent laboratory abnormalities and treatment-emergent Grade 3 or 4 laboratory abnormalities summary tables and listings:

| Battery | Lab Test Label<br>Used in I-labtox Listing | Toxicity<br>Direction | Lab Test Label<br>Used in t-labtox Table |
|---|---|---|---|
| | Hemoglobin | Decrease | Hemoglobin (Decreased) |
| II | Neutrophils | Decrease | Neutrophils (Decreased) |
| Hematology | Platelets | Decrease | Platelets (Decreased) |
| | WBC | Decrease | WBC (Decreased) |
| | Albumin | Decrease | Albumin (Decreased) |
| | Alkaline Phosphatase | Increase | Alkaline Phosphatase (Increased) |
| | ALT | Increase | ALT (Increased) |
| | Amylase | Increase | Amylase (Increased) |
| | AST | Increase | AST (Increased) |
| | Bicarbonate | Decrease | Bicarbonate (Decreased) |
| | Corrected Calcium | Increase | Corrected Calcium (Hypercalcemia) |
| | Corrected Calcium | Decrease | Corrected Calcium (Hypocalcemia) |
| | Creatine Kinase (CK) | Increase | Creatine Kinase (Increased) |
| | Creatinine | Increase | Creatinine (Increased) |
| | GGT | Increase | GGT (Increased) |
| | Lipase | Increase | Lipase (Increased) |
| | Magnesium | Decrease | Magnesium (Hypomagnesemia) |
| | Phosphate | Decrease | Phosphate (Hypophosphatemia) |
| | Serum Glucose (Fasting) | Increase | Serum Glucose (Fasting, Hyperglycemia) |
| Clara interna | Serum Glucose (Fasting) | Decrease | Serum Glucose (Fasting, Hypoglycemia) |
| Chemistry | Serum Glucose (Nonfasting) | Increase | Serum Glucose (Nonfasting, Hyperglycemia) |
| | Serum Glucose (Nonfasting) | Decrease | Serum Glucose (Nonfasting, Hypoglycemia) |
| | Serum Potassium | Increase | Serum Potassium (Hyperkalemia) |
| | Serum Potassium | Decrease | Serum Potassium (Hypokalemia) |
| | Serum Sodium | Increase | Serum Sodium (Hypernatremia) |
| | Serum Sodium | Decrease | Serum Sodium (Hyponatremia) |
| | Total Bilirubin | Increase | Total Bilirubin (Hyperbilirubinemia) |
| | Total Cholesterol (Fasting) | Increase | Total Cholesterol (Fasting, Hypercholesterolemia) |
| | Triglycerides (Fasting) | Increase | Triglycerides (Fasting, Increased) |
| | LDL (Fasting) | Increase | LDL (Fasting, Increased) |
| | Urea Nitrogen (BUN) | Increase | Urea Nitrogen (Increased) |
| | Uric Acid | Increase | Uric Acid (Hyperuricemia) |
| | Uric Acid | Decrease | Uric Acid (Hypouricemia) |
| | Prothrombin Intl. Normalized Ratio (INR) | Increase | N/A |
| | Prothrombin Time (PT) | Increase | N/A |
| | Urine Blood | Increase | N/A |
| TT: 1 : | Urine Glucose | Increase | Urine Glucose (Glycosuria) |
| Urinalysis | Urine Protein | Increase | Urine Protein (Proteinuria) |
| | Urine RBC | Increase | Urine RBC (Hematuria, Quantitative) |

Note: Prothrombin Intl. Normalized Ratio (INR) and Prothrombin Time (PT) were graded based on the protocol defined toxicity grade scale. The results and toxicity grade will be listed in listing, but not be summarized in lab toxicity summary table.

- 17) Clarification for "Pharmacokinetic Blood Sampling Time Record" listing
  - A new variable "Sample age" will be added in this listing, defined as the duration in day between sample collection date and assay date, ie, sample age = assay date sample collection date + 1.
  - SAMTIME (hours) = sample collection time (xx:xx) last dose time before sample collection (xx:xx).

Except for SAMTIME for intensive PK samples at predose:

SAMTIME (hours) = predose sample collection time (xx:xx) - dose time after predose sample collection (xx:xx).

- 18) PK parameters at the individual subject level should be displayed with the following reported number of decimal places:
  - LambdaZ, r2, r2 adj, and CORRXY: 3 decimal places
  - t<sub>1/2</sub>, T<sub>last</sub>, T<sub>max</sub>, BEGHOUR, and ENDHOUR: 2 decimal places
  - AUC<sub>tau</sub>, AUC<sub>0-last</sub>, AUC<sub>inf</sub>, %otAUC<sub>exp</sub>, Vz/F, CL/F, CLss/F, C<sub>max</sub>, C<sub>last</sub> and C<sub>tau</sub>: 1 decimal place
  - NPOINTS: 0 decimal place
  - PK concentration data will be reported with 1 decimal place.
- 19) PK parameters included in PK summary tables are defined in PK aberration listing on Page 9, except that TAF Ctau will not be included in corresponding PK summary table, since TAF Ctau should be BLQ for all subjects due to the short half-life of TAF.
  - PK parameters should be displayed as alphabetic order as listed in PK abbreviation listing.
  - SDTM.PP.PPSPID should be used as the label for each PK parameter, which also listed in PK abbreviation listing.
- 20) Concomitant nonstudy-drug ARV medications (ie, ARV medications other than study drug that are taken while receiving study drug) will be flagged in "Nonstudy-Drug Antiviral Medication" listing. The logic to define concomitant nonstudy-drug ARV is similar to concomitant non-ARV Medications (see details in Section 7.4.2)

# 21) Lipid modifying medication analyses:

- Lipid modifying medication is defined to be the concomitant medication with CMCLAS = "LIPID MODIFYING AGENTS" and CMDECOD contains wording of "STATIN" in the ADCM dataset.
- Subjects who took lipid modifying medications at study entry refer to the subjects who use of the lipid modifying agents at study day 1 (ie, the first dose date). More specifically, subjects with "Lipid Modifying Agent Use at Study Entry" include those subjects in safety analysis set with: 1) any selected CM record with the start date ≤ the first dose date, and 2) the end date of the selected CM record is ongoing or the end date of the selected CM record ≥ the first dose date.
- Subjects who initiated lipid modifying medications during the study include the subjects in the safety analysis set who didn't take lipid modifying medications at study entry and met the following criteria: 1) for subjects who permanently discontinued study drug with any selected CM record started after the first dose date and on and prior to the last dose date; 2) for subjects who are still on study drug with any selected CM records started after the first dose date.
- For lipid modifying medications with the start date completely unknown, we assume the start date is on or before the first dose date, lipid modifying medication was considered as being taken at study entry if the end date is not prior to the first dose date (ie, the end date is on or after the first dose date, completely unknown, or ongoing).
- Lipid modifying medications with the start date prior to the first dose date and the end date completely unknown were considered as being taken at study entry.
- 22) For figures, if at a visit where n (sample size) for any treatment group ≤ 5, data for that treatment group will not be displayed at the visit in figure (except the Kaplan-Meier figure), but all data will be included in the corresponding table summary.

# 23) HIV/HBV and HIV/HCV Coinfection:

• The following table presents the HBV and HCV tests with all possible values. Values that have an asterisk after them denote a "positive" (or "quantifiable" for HBV DNA and HCV RNA) result while all others denote a "negative" result.

| Label | LBTESTCD | LBTEST | Possible Values |
|---|---|---|---|
| HBsAg | CNT63 | Hep B Surface Ag | "Positive"*, "Positive, Confirmed"*, "Negative" |
| HBsAg | ATT2 | Hep. B Surf. Ag Qual(-70)-PS | "Repeat reactive, confirmed"*, "Repeat Reactive Unconfirmed", "Non-Reactive" |
| HBsAb | CNT353 | anti-Hep B Surface Ag2 Qual | "Positive"*, "Negative" |
| HBcAb | CNT68 | Hepatitis B Core Total | "Positive"*, "Negative" |
| HBV DNA | GET1883 | HBV DNA CAP/CTM<br>2.0-EDTA-CL | "No HBV DNA detected", "<20 IU/mL HBV DNA detected", ">170000000"*, NUMERICAL VALUE* |
| HCVAb | CNT350 | Hepatitis C Virus Antibody | "Positive"*, "Indeterminate", "Negative" |
| HCV RNA | GET1881 | HCV RNA CAP/CTM<br>2.0EDTA-CL | "No HCV RNA detected", "<15 IU/mL HCV RNA detected", NUMERICAL VALUE* |

- For baseline coinfection, when considering the different laboratory tests, take the latest, non-missing record on or prior to the first dose date for each test (eg, HBsAg, HBsAb, HBcAb, and HBV DNA)
  - The baseline coinfection status will be one of the three values: Yes/No/Null
  - The following tables provide combinations of HBV and HCV tests and the corresponding baseline coinfection status

| HBsAg | HBsAb | HBcAb | HBV DNA | <b>Coinfection Status</b> |
|---|---|---|---|---|
| Positive | - | - | - | Y |
| Negative | Positive | - | - | N |
| | | Positive | Quantifiable | Y |
| | | | Not Quantifiable | N |
| | | | Missing | Null |
| | Negative | Negative | - | N |
| | | Missing | Quantifiable | Null |
| | | | Not Quantifiable | N |
| | | | Missing | Null |
| | | Positive | Quantifiable | Null |
| | Missing | | Not Quantifiable | N |
| | | | Missing | Null |
| | | Negative | - | N |
| | | Missing | Quantifiable | Null |
| | | | Not Quantifiable | N |
| | | | Missing | Null |
| | Positive | - | - | Null |
| Missing | Negative | Positive | Quantifiable | Y |
| | | | Not Quantifiable | Null |
| | | | Missing | Null |
| | | Negative | - | Null |
| | | Missing | - | Null |
| | Missing | - | - | Null |

| HCVAb | HCV RNA | Coinfection Status |
|----------|------------------|--------------------|
| | Quantifiable | Y |
| Positive | Not Quantifiable | N |
| | Missing | Null |
| Negative | - | N |
| | Quantifiable | Null |
| Missing | Not Quantifiable | N |
| | Missing | Null |

<sup>&</sup>quot;-" means any value can be present, as it does not affect the classification

- For incident coinfection, all laboratory tests must share the same accession number and if any set of values meets the criteria, then the subject is considered to have incident coinfection
  - The incident coinfection status will be one of two values: Yes/Null
  - The following tables provide combinations of HBV and HCV tests that are considered "Y" for incident coinfection status (all others are considered Null)

| HBsAg | HBsAb | HBcAb | HBV DNA | <b>Coinfection Status</b> |
|----------|----------|----------|--------------|---------------------------|
| Positive | - | - | - | Y |
| Negative | Negative | Positive | Quantifiable | Y |
| Missing | Negative | Positive | Quantifiable | Y |

| HCVAb | HCV RNA | Coinfection Status |
|-----------|--------------|--------------------|
| Positive* | - | Y |
| - | Quantifiable | Y |

<sup>\*</sup> Subjects with positive HCVAb postbaseline must also have negative or missing HCVAb at baseline in order to be considered as having incident HIV/HCV coinfection.

- For adverse events, the start date must be after the first dose date and on or prior to the last dose date
- For incomplete AE start dates, please follow the logic specified in Section 7.1.5.2, but modify the second criterion to read, "The month and year (or year) of the AE onset is the same as or before the month and year (or year) of the date of the last dose of study drug".
- 24) HBV DNA test codes: If the result of the lab test code GET1883 (HBV DNA CAP/CTM 2.0-EDTA-CL) is listed as ">170000000", then a reflexive test code GET1884 (HBV DNA CAP/CTM 2.0Dil-EDTA-CL) should be performed and will share the same accession number as the original GET1883 test. In this instance, use the result from GET1884 instead of GET1883 when determining HBV DNA.

<sup>&</sup>quot;-" means any value can be present, as it does not affect the classification